CLINICAL TRIAL: NCT02954354
Title: A Phase 3, Multicenter, Randomized, Double-blind Study of a Single Dose of S-033188 (Baloxavir Marboxil) Compared With Placebo or Oseltamivir 75 mg Twice Daily for 5 Days in Otherwise Healthy Patients With Influenza
Brief Title: A Study of S-033188 (Baloxavir Marboxil) Compared With Placebo or Oseltamivir in Otherwise Healthy Patients With Influenza
Acronym: CAPSTONE 1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shionogi (Industry)
Responsible Party: Sponsor
Organization: Shionogi Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1601T0831
Record Dates: First submitted 2016-10-27; First posted 2016-11-03 (Estimated); Results first posted 2018-12-14 (Actual); Last update posted 2019-05-08 (Actual); Status verified 2019-04

CONDITIONS: Influenza
Keywords: Flu; Baloxavir Marboxil; Oseltamivir; Tamiflu®
MeSH Terms: conditions — Influenza, Human | interventions — baloxavir; Oseltamivir

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- Adults: Baloxavir Marboxil (Experimental): Participants aged 20 to 64 years will receive two or four 20 mg baloxavir marboxil tablets orally on Day 1 and one oseltamivir placebo capsule orally twice a day (BID) on Days 1 to 5.
  Interventions: Drug: Baloxavir Marboxil; Drug: Placebo to Oseltamivir
- Adults: Oseltamivir (Active Comparator): Participants aged 20 to 64 years will receive 75 mg oseltamivir twice a day on Days 1 to 5 and two or four baloxavir marboxil placebo tablets on Day 1.
  Interventions: Drug: Placebo to Baloxavir Marboxil; Drug: Oseltamivir
- Adults: Placebo (Placebo Comparator): Participants aged 20 to 64 years will receive two or four baloxavir marboxil placebo tablets on Day 1 and one oseltamivir placebo capsule orally twice a day on Days 1 to 5.
  Interventions: Drug: Placebo to Baloxavir Marboxil; Drug: Placebo to Oseltamivir
- Adolescents: Baloxavir Marboxil (Experimental): Participants aged 12 to 19 years will receive two or four baloxavir marboxil 20 mg tablets on Day 1.
  Interventions: Drug: Baloxavir Marboxil
- Adolescents: Placebo (Placebo Comparator): Participants aged 12 to 19 years will receive two or four baloxavir marboxil placebo tablets on Day 1.
  Interventions: Drug: Placebo to Baloxavir Marboxil

INTERVENTIONS:
Drug: Baloxavir Marboxil — 2 to4 X 20-mg tablets taken orally
  Other Names: S-033188
  Arms: Adolescents: Baloxavir Marboxil; Adults: Baloxavir Marboxil
Drug: Placebo to Baloxavir Marboxil — 2 to4 X 20-mg tablets taken orally
  Arms: Adolescents: Placebo; Adults: Oseltamivir; Adults: Placebo
Drug: Oseltamivir — 75 mg capsules taken orally
  Other Names: Tamiflu®
  Arms: Adults: Oseltamivir
Drug: Placebo to Oseltamivir — Placebo capsules matching oseltamivir 75 mg capsules
  Arms: Adults: Baloxavir Marboxil; Adults: Placebo

SUMMARY:
The primary objective of this study is to evaluate the efficacy of a single, oral dose of baloxavir marboxil compared with placebo by measuring the time to alleviation of symptoms in patients with uncomplicated influenza virus infection.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who are able to understand the study and comply with all study procedures, and willing to provide written informed consent/assent prior to the predose examinations appropriately. As for adolescent patients, informed consent/assent of voluntary participation should be obtained in accordance with local requirements
2. Male or female patients aged ≥ 12 to ≤ 64 years at the time of signing the informed consent/assent form.
3. Patients with a diagnosis of influenza virus infection confirmed by all of the following:

   1. Fever ≥ 38ºC (axillary) in the predose examinations or > 4 hours after dosing of antipyretics if they were taken
   2. At least one of the following general systemic symptoms associated with influenza are present with a severity of moderate or greater

      * Headache
      * Feverishness or chills
      * Muscle or joint pain
      * Fatigue
   3. At least one of the following respiratory symptoms associated with influenza are present with a severity of moderate or greater

      * Cough
      * Sore throat
      * Nasal congestion
4. The time interval between the onset of symptoms and the predose examinations is 48 hours or less. The onset of symptoms is defined as either:

   1. Time of the first increase in body temperature (an increase of at least 1ºC from normal body temperature)
   2. Time when the patient experiences at least one general or respiratory symptom
5. Women of childbearing potential who agree to use a highly effective method of contraception for 3 months after the first dose of study drug

Exclusion Criteria:

1. Patients with severe influenza virus infection requiring inpatient treatment.
2. Patients aged ≥ 20 years with known allergy to oseltamivir (Tamiflu®).
3. Patients with any of the following risk factors

   1. Women who are pregnant or within 2 weeks post-partum
   2. Residents of long-term care facilities (eg, welfare facilities for the elderly, nursing homes)
   3. Chronic respiratory diseases including bronchial asthma
   4. Neurological and neurodevelopmental disorders including disorders of the brain, spinal cord, peripheral nerve, and muscle (eg, cerebral palsy, epilepsy [seizure disorders], stroke, intellectual disability, moderate to severe developmental delay, muscular dystrophy, or spinal cord injury)
   5. Heart disease (such as congenital heart disease, congestive heart failure, or coronary artery disease), excluding hypertension without any other heart-related symptoms)
   6. American Indians and Alaskan natives
   7. Blood disorders (such as sickle cell disease)
   8. Endocrine disorders (including diabetes mellitus)
   9. Kidney disorders
   10. Liver disorders
   11. Metabolic disorders
   12. Compromised immune system (including patients receiving immunosuppressant therapy, or those with cancer or human immunodeficiency virus [HIV] infection)
   13. Morbid obesity (body mass index [BMI] ≥ 40)
4. Patients unable to swallow tablets or capsules.
5. Patients who have previously received Baloxavir Marboxil.
6. Patients weighing < 40 kg
7. Patients who have been exposed to an investigational drug within 30 days prior to the predose examinations.
8. Women who are breastfeeding or have a positive pregnancy test in the predose examinations. The following female patients who have documentation of either a or b below do not need to undergo a pregnancy test in the predose examinations:

   1. Postmenopausal (defined as cessation of regular menstrual periods for 2 years or more and confirmed by a follicle-stimulating hormone test) women
   2. Women who are surgically sterile by hysterectomy, bilateral oophorectomy, or tubal ligation
9. Patients with concurrent infections requiring systemic antimicrobial and/or antiviral therapy at the predose examinations.
10. Patients who have received peramivir, laninamivir, oseltamivir, zanamivir, rimantadine, umifenovir, or amantadine within 30 days prior to the predose examinations.
11. Patients who have received an investigational monoclonal antibody for a viral disease in the last year.
12. Patients with severe underlying diseases.
13. Patients with known creatinine clearance ≤ 60 mL/min.
14. Patients who, in the opinion of the investigator, would be unlikely to comply with required study visits, self-assessments, and interventions

Ages: 12 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1436 (Actual)
Dates: Start 2016-12-08 (Actual); Primary Completion 2017-04-04 (Actual); Study Completion 2017-04-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Support Help Line Shionogi Clinical Trials Administrator, Study Director — Shionogi

REFERENCES:
- [Result] Hayden FG, Sugaya N, Hirotsu N, Lee N, de Jong MD, Hurt AC, Ishida T, Sekino H, Yamada K, Portsmouth S, Kawaguchi K, Shishido T, Arai M, Tsuchiya K, Uehara T, Watanabe A; Baloxavir Marboxil Investigators Group. Baloxavir Marboxil for Uncomplicated Influenza in Adults and Adolescents. N Engl J Med. 2018 Sep 6;379(10):913-923. doi: 10.1056/NEJMoa1716197. PMID 30184455
- [Derived] Retout S, De Buck S, Jolivet S, Duval V, Cosson V. A Pharmacokinetics-Time to Alleviation of Symptoms Model to Support Extrapolation of Baloxavir Marboxil Clinical Efficacy in Different Ethnic Groups with Influenza A or B. Clin Pharmacol Ther. 2022 Aug;112(2):372-381. doi: 10.1002/cpt.2648. Epub 2022 Jun 10. PMID 35585696
- [Derived] Uehara T, Hayden FG, Kawaguchi K, Omoto S, Hurt AC, De Jong MD, Hirotsu N, Sugaya N, Lee N, Baba K, Shishido T, Tsuchiya K, Portsmouth S, Kida H. Treatment-Emergent Influenza Variant Viruses With Reduced Baloxavir Susceptibility: Impact on Clinical and Virologic Outcomes in Uncomplicated Influenza. J Infect Dis. 2020 Jan 14;221(3):346-355. doi: 10.1093/infdis/jiz244. PMID 31309975

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 297 sites, consisting of 141 sites in Japan, 149 sites in the United States, and 7 sites in Canada. Participants were enrolled from December 2016 to April 2017.
Pre-assignment Details: Participants 20 to 64 years of age were randomly assigned in a 2:2:1 ratio to receive a single oral dose of baloxavir, 75 mg oseltamivir twice daily for 5 days, or matching placebos.
  Participants 12 to 19 years of age were randomly assigned in a 2:1 ratio to receive a single dose of either baloxavir or placebo.
Groups:
- Baloxavir: Participants aged 20 to 64 years received 40 mg or 80 mg baloxavir (depending on weight) orally on Day 1 and placebo to oseltamivir orally twice a day (BID) on Days 1 to 5.
  Participants aged 12 to 19 years received 40 mg or 80 mg baloxavir (depending on weight) on Day 1.
- Placebo: Participants aged 20 to 64 years received placebo to baloxavir on Day 1 and placebo to oseltamivir orally twice a day on Days 1 to 5. Participants aged 12 to 19 years received placebo to baloxavir on Day 1.
- Oseltamivir: Participants aged 20 to 64 years received 75 mg oseltamivir orally BID on Days 1 to 5 and placebo to baloxavir on Day 1.
Period: Overall Study
Arm/Group | Baloxavir | Placebo | Oseltamivir
Started | 612 | 310 | 514
Received Study Drug | 610 | 309 | 513
Intention to Treat Infected Population | 456 | 231 | 377
Completed | 578 | 290 | 498
Not Completed | 34 | 20 | 16
Not completed — Adverse Event | 2 | 2 | 4
Not completed — Failure to Meet Eligibility Criteria | 1 | 0 | 0
Not completed — Lack of Efficacy | 0 | 2 | 0
Not completed — Withdrawal by Subject | 17 | 9 | 11
Not completed — Lost to Follow-up | 12 | 5 | 0
Not completed — Miscellaneous | 2 | 2 | 1

BASELINE CHARACTERISTICS:
Population: Intention-to-treat infection (ITTI) population consisting of participants who received study drug with a confirmed diagnosis of influenza. Confirmation of influenza was based on the results of reverse transcription polymerase chain reaction (RT-PCR) on Day 1.
Groups:
- Total: Total of all reporting groups
Arm/Group | Baloxavir | Placebo | Oseltamivir | Total
Number analyzed (Participants) | 456 | 231 | 377 | 1064
Age, Continuous [Mean (Standard Deviation); unit: Years] — Note that the baloxavir and placebo groups included participants from 12 to 64 years of age whereas the oseltamivir group only included participants from 20 to 64 years of age.
  Years | 33.5 (13.5) | 33.9 (13.7) | 36.0 (11.8) | 34.5 (13.0)
Age, Customized [Count of Participants; unit: Participants]
  ≥ 12 to ≤ 19 years | 80 | 38 | 0 | 118
  ≥ 20 to ≤ 29 years | 121 | 61 | 134 | 316
  ≥ 30 to ≤ 39 years | 92 | 47 | 104 | 243
  ≥ 40 to ≤ 49 years | 97 | 48 | 77 | 222
  ≥ 50 to ≤ 59 years | 52 | 30 | 51 | 133
  ≥ 60 to ≤ 64 years | 14 | 7 | 11 | 32
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 224 | 111 | 159 | 494
  Male | 232 | 120 | 218 | 570
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 32 | 11 | 25 | 68
  Not Hispanic or Latino | 424 | 220 | 352 | 996
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 349 | 178 | 305 | 832
  Black or African American | 18 | 11 | 9 | 38
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 1
  White | 85 | 40 | 60 | 185
  Other | 4 | 2 | 2 | 8
Time From Symptom Onset to Initiation of the Trial Regimen [Count of Participants; unit: Participants]
  ≥ 0 to ≤ 12 hours | 60 | 34 | 41 | 135
  > 12 to ≤ 24 hours | 178 | 87 | 163 | 428
  > 24 to ≤ 36 hours | 139 | 67 | 94 | 300
  > 36 to ≤ 48 hours | 79 | 43 | 79 | 201
Influenza Virus Type or Subtype on RT-PCR Assay at Enrollment [Count of Participants; unit: Participants]
  A/H1N1pdm | 7 | 7 | 2 | 16
  A/H3 | 393 | 196 | 332 | 921
  B | 38 | 20 | 34 | 92
  Mixed infection | 8 | 3 | 6 | 17
  Other | 10 | 5 | 3 | 18
Region [Count of Participants; unit: Participants]
  Japan/Asia | 343 | 175 | 303 | 821
  Rest of the world | 113 | 56 | 74 | 243
Composite Symptom Score [Count of Participants; unit: Participants] — Participants assessed the severity of seven influenza-associated symptoms (cough, sore throat, headache, nasal congestion, feverishness or chills, muscle or joint pain, and fatigue) on a 4-point scale (with 0 indicating no symptoms, 1 mild symptoms, 2 moderate symptoms, and 3 severe symptoms). The composite symptom score is the total score of the 7 influenza symptoms as assessed by the participant, and ranges from 0 to 21.
  Participants
    ≤ 11 | 144 | 72 | 119 | 335
    ≥ 12 | 312 | 159 | 258 | 729

OUTCOME MEASURES:

1. Primary Outcome: Time to Alleviation of Symptoms in Participants Randomized to Baloxavir or Placebo
Description: Participants assessed the severity of seven influenza-associated symptoms (cough, sore throat, headache, nasal congestion, feverishness or chills, muscle or joint pain, and fatigue) on a 4-point scale (with 0 indicating no symptoms, 1 mild symptoms, 2 moderate symptoms, and 3 severe symptoms).
  Time to alleviation of symptoms was defined as the time from the start of the study treatment to the time when all seven influenza-related symptoms were assessed by the participant as absent (0) or mild (1) for at least 21.5 hours.
  Time to alleviation of symptoms was analyzed using the Kaplan-Meier (KM) method; participants who did not experience alleviation of symptoms were censored at the last observation time point.
Time Frame: Initiation of study treatment up to Day 14
Population: Participants in the intention-to-treat infection population assigned to baloxavir or placebo with available time to alleviation of symptoms data.
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | Baloxavir | Placebo
Number analyzed (Participants) | 455 | 230
hours | 53.7 [49.5 to 58.5] | 80.2 [72.6 to 87.1]
Statistical Analysis 1: Comparison: Baloxavir vs Placebo; The primary analysis of time to alleviation of symptoms was a comparison of baloxavir with placebo in all participants in the intention-to-treat infection population. Statistical tests were performed at the 0.05 significance level; Test type: Superiority; p < 0.0001, Generalized Wilcoxon test — Adjusted p-value, two-sided significance level of 0.05; Generalized Wilcoxon test stratified by composite symptom scores at baseline (≤ 11 or ≥ 12) and region (Japan/Asia or Rest of the world); Difference = -26.5, 95% CI 2-sided [-35.8 to -17.8]
Statistical Analysis 2: Comparison: Baloxavir vs Placebo; Analysis using the stratified log rank test was performed as a sensitivity analysis; Test type: Superiority; p < 0.0001, Log Rank — The p-value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; Log rank test stratified by composite symptom scores at baseline (≤ 11 or ≥ 12) and region (Japan/Asia or Rest of the world)

2. Primary Outcome: Time to Alleviation of Symptoms in Adults Randomized to Baloxavir or Oseltamivir
Description: Participants assessed the severity of seven influenza-associated symptoms (cough, sore throat, headache, nasal congestion, feverishness or chills, muscle or joint pain, and fatigue) on a 4-point scale (with 0 indicating no symptoms, 1 mild symptoms, 2 moderate symptoms, and 3 severe symptoms).
  Time to alleviation of symptoms was defined as the time from the start of the study treatment to the time when all seven influenza-related symptoms were assessed by the participant as absent (0) or mild (1) for at least 21.5 hours.
  Time to alleviation of symptoms was analyzed using the Kaplan-Meier(KM) method; participants who did not experience alleviation of symptoms were censored at the last observation time point.
Time Frame: Initiation of study treatment up to Day 14
Population: Participants in the intention-to-treat infection population, ≥ 20 years of age and assigned to baloxavir or oseltamivir, and with available time to alleviation of symptoms data.
Measure: Median (95% Confidence Interval); unit: hours
Groups:
- Baloxavir: Participants aged 20 to 64 years received 40 mg or 80 mg baloxavir (depending on weight) orally on Day 1 and placebo to oseltamivir orally twice a day (BID) on Days 1 to 5.
Arm/Group | Baloxavir | Oseltamivir
Number analyzed (Participants) | 375 | 377
hours | 53.5 [48.0 to 58.5] | 53.8 [50.2 to 56.4]
Statistical Analysis 1: Comparison: Baloxavir vs Oseltamivir; A secondary analysis of time to alleviation of symptoms, consisting of a comparison between the 20 to 64 years of age stratum of the baloxavir group and the oseltamivir group, was conducted if statistical significance was observed in the primary analysis in order to maintain the overall Type I error; Test type: Superiority; p = 0.7560, Generalized Wilcoxon test — Adjusted p-value, two-sided significance level of 0.05; [statistical method as in outcome 1, analysis 1]; Difference = -0.3, 95% CI 2-sided [-6.6 to 6.6]
Statistical Analysis 2: Comparison: Baloxavir vs Oseltamivir; Analysis using the stratified log rank test was performed as a sensitivity analysis; Test type: Superiority; p = 0.3761, Log Rank — The p-value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 1, analysis 2]

3. Secondary Outcome: Percentage of Participants With Positive Influenza Virus Titer at Each Time Point in Participants Randomized to Baloxavir or Placebo
Description: Virus titer was quantified from nasopharyngeal swabs (or throat swabs if nasopharyngeal swabbing was not feasible) by tissue culture methods. Positive influenza virus titer was defined as virus titer not less than the lower limit of quantification (0.7 log₁₀ of the 50% tissue culture infective dose (TCID₅₀/mL) among those assessed for virus titer on Days 2, 3, 4, 5, 6 and 9.
Time Frame: Days 2, 3, 4 (optional), 5, 6 (optional), and 9
Population: Participants in the intention-to-treat infection population assigned to baloxavir or placebo, with positive influenza virus titer on Day 1 and with available virus titer data at each time point.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Baloxavir | Placebo
Number analyzed (Participants) | 427 | 210
percentage of participants
  Day 2: number analyzed (Participants) | 414 | 201
  Day 2 | 47.6 [42.7 to 52.5] | 96.0 [92.3 to 98.3]
  Day 3: number analyzed (Participants) | 406 | 193
  Day 3 | 21.7 [17.8 to 26.0] | 70.5 [63.5 to 76.8]
  Day 4: number analyzed (Participants) | 114 | 57
  Day 4 | 16.7 [10.3 to 24.8] | 56.1 [42.4 to 69.3]
  Day 5: number analyzed (Participants) | 406 | 192
  Day 5 | 13.5 [10.4 to 17.3] | 29.7 [23.3 to 36.7]
  Day 6: number analyzed (Participants) | 97 | 48
  Day 6 | 8.2 [3.6 to 15.6] | 12.5 [4.7 to 25.2]
  Day 9: number analyzed (Participants) | 408 | 197
  Day 9 | 2.9 [1.5 to 5.1] | 4.6 [2.1 to 8.5]
Statistical Analysis 1: Comparison: Baloxavir vs Placebo; Day 2; Test type: Superiority; p < 0.0001, Mantel Haenszel — The p-value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; Mantel-Haenszel test stratified by composite symptom scores at baseline (≤ 11 or ≥ 12) and region (Japan/Asia or Rest of the world)
Statistical Analysis 2: Comparison: Baloxavir vs Placebo; Day 3; Test type: Superiority; p < 0.0001, Mantel Haenszel — The p-value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 3, analysis 1]
Statistical Analysis 3: Comparison: Baloxavir vs Placebo; Day 4; Test type: Superiority; p < 0.0001, Mantel Haenszel — The p-value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 3, analysis 1]
Statistical Analysis 4: Comparison: Baloxavir vs Placebo; Day 5; Test type: Superiority; p < 0.0001, Mantel Haenszel — The p-value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 3, analysis 1]
Statistical Analysis 5: Comparison: Baloxavir vs Placebo; Day 6; Test type: Superiority; p = 0.4767, Mantel Haenszel — The p-value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 3, analysis 1]
Statistical Analysis 6: Comparison: Baloxavir vs Placebo; Day 9; Test type: Superiority; p = 0.3353, Mantel Haenszel — The p-value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 3, analysis 1]

4. Secondary Outcome: Percentage of Participants With Positive Influenza Virus Titer at Each Time Point in Adults Randomized to Baloxavir or Oseltamivir
Description: as for outcome 3
Time Frame: Days 2, 3, 4 (optional), 5, 6 (optional), and 9
Population: Participants in the intention-to-treat infection population, ≥ 20 years of age and assigned to baloxavir or oseltamivir, with positive influenza virus titer on Day 1 and with available virus titer data at each time point.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Baloxavir | Oseltamivir
Number analyzed (Participants) | 352 | 359
percentage of participants
  Day 2: number analyzed (Participants) | 340 | 348
  Day 2 | 47.4 [41.9 to 52.8] | 91.1 [87.6 to 93.9]
  Day 3: number analyzed (Participants) | 335 | 344
  Day 3 | 20.0 [15.8 to 24.7] | 57.3 [51.9 to 62.6]
  Day 4: number analyzed (Participants) | 87 | 105
  Day 4 | 16.1 [9.1 to 25.5] | 27.6 [19.3 to 37.2]
  Day 5: number analyzed (Participants) | 333 | 336
  Day 5 | 12.9 [9.5 to 17.0] | 20.8 [16.6 to 25.6]
  Day 6: number analyzed (Participants) | 71 | 78
  Day 6 | 5.6 [1.6 to 13.8] | 9.0 [3.7 to 17.6]
  Day 9: number analyzed (Participants) | 336 | 340
  Day 9 | 3.0 [1.4 to 5.4] | 3.2 [1.6 to 5.7]
Statistical Analysis 1: Comparison: Baloxavir vs Oseltamivir; Day 2; Test type: Superiority; p < 0.0001, Mantel Haenszel — The p-value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 3, analysis 1]
Statistical Analysis 2: Comparison: Baloxavir vs Oseltamivir; Day 3; Test type: Superiority; p < 0.0001, Mantel Haenszel — The p-value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 3, analysis 1]
Statistical Analysis 3: Comparison: Baloxavir vs Oseltamivir; Day 4; Test type: Superiority; p = 0.0852, Mantel Haenszel — The p-value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 3, analysis 1]
Statistical Analysis 4: Comparison: Baloxavir vs Oseltamivir; Day 5; Test type: Superiority; p = 0.0063, Mantel Haenszel — The p-value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 3, analysis 1]
Statistical Analysis 5: Comparison: Baloxavir vs Oseltamivir; Day 6; Test type: Superiority; p = 0.6187, Mantel Haenszel — The p-value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 3, analysis 1]
Statistical Analysis 6: Comparison: Baloxavir vs Oseltamivir; Day 9; Test type: Superiority; p = 0.8637, Mantel Haenszel — The p-value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05

5. Secondary Outcome: Percentage of Participants With Positive Influenza Virus by RT-PCR at Each Time Point in Participants Randomized to Baloxavir or Placebo
Description: Influenza virus ribonucleic acid (RNA) was quantified from nasopharyngeal swabs (or throat swabs, if nasopharyngeal swabbing was not feasible). The percentage of participants with detectable virus RNA (2.05 for flu A and 2.83 for flu B log₁₀ virus particles/mL) among those assessed measured by reverse transcription polymerase chain reaction (RT-PCR) on Days 2, 3, 4, 5, 6 and 9.
Time Frame: Days 2, 3, 4 (optional), 5, 6 (optional), and 9
Population: Participants in the intention-to-treat infection population assigned to baloxavir or placebo, with positive influenza virus RNA determined by RT-PCR on Day 1 and with available data at each time point were included in the analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Baloxavir | Placebo
Number analyzed (Participants) | 456 | 231
percentage of participants
  Day 2: number analyzed (Participants) | 443 | 222
  Day 2 | 97.3 [95.3 to 98.6] | 97.7 [94.8 to 99.3]
  Day 3: number analyzed (Participants) | 436 | 214
  Day 3 | 95.6 [93.3 to 97.4] | 97.2 [94.0 to 99.0]
  Day 4: number analyzed (Participants) | 122 | 67
  Day 4 | 93.4 [87.5 to 97.1] | 91.0 [81.5 to 96.6]
  Day 5: number analyzed (Participants) | 436 | 213
  Day 5 | 87.4 [83.9 to 90.4] | 93.9 [89.8 to 96.7]
  Day 6: number analyzed (Participants) | 103 | 57
  Day 6 | 74.8 [65.2 to 82.8] | 77.2 [64.2 to 87.3]
  Day 9: number analyzed (Participants) | 436 | 217
  Day 9 | 61.5 [56.7 to 66.1] | 72.4 [65.9 to 78.2]
Statistical Analysis 1: Comparison: Baloxavir vs Placebo; Day 2; Test type: Superiority; p = 0.6145, Mantel Haenszel — The p-value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 3, analysis 1]
Statistical Analysis 2: Comparison: Baloxavir vs Placebo; Day 3; Test type: Superiority; p = 0.2505, Mantel Haenszel — The p-value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 3, analysis 1]
Statistical Analysis 3: Comparison: Baloxavir vs Placebo; Day 4; Test type: Superiority; p = 0.4190, Mantel Haenszel — The p-value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 3, analysis 1]
Statistical Analysis 4: Comparison: Baloxavir vs Placebo; Day 5; Test type: Superiority; p = 0.0095, Mantel Haenszel — The p-value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 3, analysis 1]
Statistical Analysis 5: Comparison: Baloxavir vs Placebo; Day 6; Test type: Superiority; p = 0.7393, Mantel Haenszel — The p-value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 3, analysis 1]
Statistical Analysis 6: Comparison: Baloxavir vs Placebo; Day 9; Test type: Superiority; p = 0.0049, Mantel Haenszel — The p-value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 3, analysis 1]

6. Secondary Outcome: Percentage of Participants With Positive Influenza Virus by RT-PCR at Each Time Point in Adults Randomized to Baloxavir or Oseltamivir
Description: Influenza virus RNA was quantified from nasopharyngeal swabs (or throat swabs, if nasopharyngeal swabbing was not feasible). The percentage of participants with detectable virus RNA (2.05 for flu A and 2.83 for flu B log₁₀ virus particles/mL) among those assessed measured by reverse transcription polymerase chain reaction (RT-PCR) on Days 2, 3, 4, 5, 6 and 9.
Time Frame: Days 2, 3, 4 (optional), 5, 6 (optional), and 9
Population: Participants in the intention-to-treat infection population, ≥ 20 years of age and assigned to baloxavir or oseltamivir, with positive influenza virus RNA determined by RT-PCR on Day 1, and with available data at each time point were included in the analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Baloxavir | Oseltamivir
Number analyzed (Participants) | 376 | 377
percentage of participants
  Day 2: number analyzed (Participants) | 364 | 362
  Day 2 | 97.3 [95.0 to 98.7] | 98.6 [96.8 to 99.6]
  Day 3: number analyzed (Participants) | 360 | 362
  Day 3 | 95.3 [92.5 to 97.2] | 97.5 [95.3 to 98.9]
  Day 4: number analyzed (Participants) | 94 | 115
  Day 4 | 93.6 [86.6 to 97.6] | 93.0 [86.8 to 96.9]
  Day 5: number analyzed (Participants) | 358 | 353
  Day 5 | 86.6 [82.6 to 89.9] | 92.1 [88.7 to 94.7]
  Day 6: number analyzed (Participants) | 75 | 83
  Day 6 | 69.3 [57.6 to 79.5] | 80.7 [70.6 to 88.6]
  Day 9: number analyzed (Participants) | 359 | 360
  Day 9 | 60.2 [54.9 to 65.3] | 64.7 [59.5 to 69.7]
Statistical Analysis 1: Comparison: Baloxavir vs Oseltamivir; Day 2; Test type: Superiority; p = 0.2266, Mantel Haenszel — The p-value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 3, analysis 1]
Statistical Analysis 2: Comparison: Baloxavir vs Oseltamivir; Day 3; Test type: Superiority; p = 0.1379, Mantel Haenszel — The p-value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 3, analysis 1]
Statistical Analysis 3: Comparison: Baloxavir vs Oseltamivir; Day 4; Test type: Superiority; p = 0.5479, Mantel Haenszel — The p-value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 3, analysis 1]
Statistical Analysis 4: Comparison: Baloxavir vs Oseltamivir; Day 5; Test type: Superiority; p = 0.0241, Mantel Haenszel — The p-value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 3, analysis 1]
Statistical Analysis 5: Comparison: Baloxavir vs Oseltamivir; Day 6; Test type: Superiority; p = 0.0898, Mantel Haenszel — The p-value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 3, analysis 1]
Statistical Analysis 6: Comparison: Baloxavir vs Oseltamivir; Day 9; Test type: Superiority; p = 0.2548, Mantel Haenszel — The p-value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 3, analysis 1]

7. Secondary Outcome: Change From Baseline in Virus Titer at Each Time Point in Participants Randomized to Baloxavir or Placebo
Description: Virus titer was quantified from nasopharyngeal swabs (or throat swabs if nasopharyngeal swabbing was not feasible) by tissue culture methods.
  If virus titer was less than the lower limit of quantification, the virus titer was imputed 0.7 (TCID₅₀/mL).
Time Frame: Day 1 pretreatment (Baseline) and Days 2, 3, 4 (optional), 5, 6 (optional), and 9
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: log₁₀[TCID₅₀/mL]
Arm/Group | Baloxavir | Placebo
Number analyzed (Participants) | 427 | 210
log₁₀[TCID₅₀/mL]
  Day 2: number analyzed (Participants) | 414 | 201
  Day 2 | -4.45 (2.03) | -1.19 (2.43)
  Day 3: number analyzed (Participants) | 406 | 193
  Day 3 | -4.82 (1.99) | -2.88 (2.88)
  Day 4: number analyzed (Participants) | 114 | 57
  Day 4 | -4.50 (2.02) | -3.31 (2.34)
  Day 5: number analyzed (Participants) | 406 | 192
  Day 5 | -4.95 (1.93) | -4.47 (2.21)
  Day 6: number analyzed (Participants) | 97 | 48
  Day 6 | -4.58 (1.99) | -4.68 (2.12)
  Day 9: number analyzed (Participants) | 408 | 197
  Day 9 | -5.06 (1.87) | -4.87 (1.85)
Statistical Analysis 1: Comparison: Baloxavir vs Placebo; Day 2; Test type: Superiority; p < 0.0001, van Elteren test — The p-value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; Van Elteren test stratified by composite symptom scores at baseline (≤ 11 or ≥ 12) and region (Japan/Asia or Rest of the world)
Statistical Analysis 2: Comparison: Baloxavir vs Placebo; Day 3; Test type: Superiority; p < 0.0001, van Elteren test — The p-value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 7, analysis 1]
Statistical Analysis 3: Comparison: Baloxavir vs Placebo; Day 4; Test type: Superiority; p = 0.0008, van Elteren test — The p-value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 7, analysis 1]
Statistical Analysis 4: Comparison: Baloxavir vs Placebo; Day 5; Test type: Superiority; p = 0.0132, van Elteren test — The p-value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 7, analysis 1]
Statistical Analysis 5: Comparison: Baloxavir vs Placebo; Day 6; Test type: Superiority; p = 0.9307, van Elteren test — The p-value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 7, analysis 1]
Statistical Analysis 6: Comparison: Baloxavir vs Placebo; Day 9; Test type: Superiority; p = 0.1677, van Elteren test — The p-value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 7, analysis 1]

8. Secondary Outcome: Change From Baseline in Virus Titer at Each Time Point in Adults Randomized to Baloxavir or Oseltamivir
Description: as for outcome 7
Time Frame: Day 1 pretreatment (Baseline) and Days 2, 3, 4 (optional), 5, 6 (optional), and 9
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: log₁₀[TCID₅₀/mL]
Arm/Group | Baloxavir | Oseltamivir
Number analyzed (Participants) | 352 | 359
log₁₀[TCID₅₀/mL]
  Day 2: number analyzed (Participants) | 340 | 348
  Day 2 | -4.39 (2.07) | -2.53 (2.03)
  Day 3: number analyzed (Participants) | 335 | 344
  Day 3 | -4.79 (2.03) | -4.20 (2.02)
  Day 4: number analyzed (Participants) | 87 | 105
  Day 4 | -4.46 (2.03) | -4.63 (1.89)
  Day 5: number analyzed (Participants) | 333 | 336
  Day 5 | -4.95 (1.94) | -4.98 (1.81)
  Day 6: number analyzed (Participants) | 71 | 78
  Day 6 | -4.56 (1.99) | -4.85 (1.95)
  Day 9: number analyzed (Participants) | 336 | 340
  Day 9 | -5.03 (1.89) | -5.22 (1.70)
Statistical Analysis 1: Comparison: Baloxavir vs Oseltamivir; Day 2; Test type: Superiority; p < 0.0001, van Elteren test — The p-value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 7, analysis 1]
Statistical Analysis 2: Comparison: Baloxavir vs Oseltamivir; Day 3; Test type: Superiority; p < 0.0001, van Elteren test — The p-value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 7, analysis 1]
Statistical Analysis 3: Comparison: Baloxavir vs Oseltamivir; Day 4; Test type: Superiority; p = 0.8010, van Elteren test — The p-value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 7, analysis 1]
Statistical Analysis 4: Comparison: Baloxavir vs Oseltamivir; Day 5; Test type: Superiority; p = 0.9451, van Elteren test — The p-value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 7, analysis 1]
Statistical Analysis 5: Comparison: Baloxavir vs Oseltamivir; Day 6; Test type: Superiority; p = 0.2256, van Elteren test — The p-value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 7, analysis 1]
Statistical Analysis 6: Comparison: Baloxavir vs Oseltamivir; Day 9; Test type: Superiority; p = 0.3332, van Elteren test — The p-value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 7, analysis 1]

9. Secondary Outcome: Change From Baseline in Virus RNA (RT-PCR) at Each Time Point in Participants Randomized to Baloxavir or Placebo
Description: Nasopharyngeal swabs (or throat swabs, if nasopharyngeal swabbing was not feasible) were obtained for viral quantitation. Virus RNA is measured by reverse transcription polymerase chain reaction (RT-PCR).
Time Frame: Day 1 pretreatment (Baseline) and Days 2, 3, 4 (optional), 5, 6 (optional), and 9
Population: Participants in the intention-to-treat infection population assigned to baloxavir or placebo, with positive influenza virus titer on Day 1 and with available virus RNA data at each time point.
Measure: Mean (Standard Deviation); unit: log₁₀ virus particles/mL
Arm/Group | Baloxavir | Placebo
Number analyzed (Participants) | 456 | 231
log₁₀ virus particles/mL
  Day 2: number analyzed (Participants) | 431 | 213
  Day 2 | -1.63 (1.03) | -0.56 (1.37)
  Day 3: number analyzed (Participants) | 424 | 205
  Day 3 | -2.80 (1.20) | -1.61 (1.76)
  Day 4: number analyzed (Participants) | 120 | 66
  Day 4 | -3.07 (1.59) | -1.95 (1.76)
  Day 5: number analyzed (Participants) | 424 | 204
  Day 5 | -3.75 (1.47) | -3.04 (1.62)
  Day 6: number analyzed (Participants) | 101 | 56
  Day 6 | -3.83 (1.64) | -3.03 (1.85)
  Day 9: number analyzed (Participants) | 426 | 208
  Day 9 | -4.43 (1.42) | -4.06 (1.47)
Statistical Analysis 1: Comparison: Baloxavir vs Placebo; Day 2; Test type: Superiority; p < 0.0001, van Elteren test — The p-value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 7, analysis 1]
Statistical Analysis 2: Comparison: Baloxavir vs Placebo; Day 3; Test type: Superiority; p < 0.0001, van Elteren test — The p-value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 7, analysis 1]
Statistical Analysis 3: Comparison: Baloxavir vs Placebo; Day 4; Test type: Superiority; p < 0.0001, van Elteren test — The p-value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 7, analysis 1]
Statistical Analysis 4: Comparison: Baloxavir vs Placebo; Day 5; Test type: Superiority; p < 0.0001, van Elteren test — The p-value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 7, analysis 1]
Statistical Analysis 5: Comparison: Baloxavir vs Placebo; Day 6; Test type: Superiority; p = 0.0010, van Elteren test — The p-value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 7, analysis 1]
Statistical Analysis 6: Comparison: Baloxavir vs Placebo; Day 9; Test type: Superiority; p = 0.0002, van Elteren test — The p-value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 7, analysis 1]

10. Secondary Outcome: Change From Baseline in Virus RNA (RT-PCR) at Each Time Point in Adults Randomized to Baloxavir or Oseltamivir
Description: Nasopharyngeal swabs (or throat swabs, if nasopharyngeal swabbing was not feasible) were obtained for viral quantitation. Virus RNA was measured by reverse transcription polymerase chain reaction (RT-PCR).
Time Frame: Day 1 pretreatment (Baseline) and Days 2, 3, 4 (optional), 5, 6 (optional), and 9
Population: Participants in the intention-to-treat infection population ≥ 20 years of age and assigned to baloxavir or oseltamivir, with positive influenza virus titer on Day 1 and with available virus RNA data at each time point.
Measure: Mean (Standard Deviation); unit: log₁₀ virus particles/mL
Arm/Group | Baloxavir | Oseltamivir
Number analyzed (Participants) | 376 | 377
log₁₀ virus particles/mL
  Day 2: number analyzed (Participants) | 355 | 354
  Day 2 | -1.61 (1.06) | -1.10 (1.10)
  Day 3: number analyzed (Participants) | 350 | 352
  Day 3 | -2.79 (1.21) | -2.44 (1.24)
  Day 4: number analyzed (Participants) | 92 | 112
  Day 4 | -2.94 (1.62) | -2.97 (1.29)
  Day 5: number analyzed (Participants) | 348 | 343
  Day 5 | -3.76 (1.44) | -3.62 (1.34)
  Day 6: number analyzed (Participants) | 73 | 81
  Day 6 | -3.81 (1.52) | -3.88 (1.35)
  Day 9: number analyzed (Participants) | 351 | 349
  Day 9 | -4.43 (1.43) | -4.52 (1.22)
Statistical Analysis 1: Comparison: Baloxavir vs Oseltamivir; Day 2; Test type: Superiority; p < 0.0001, van Elteren test — The p-value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 7, analysis 1]
Statistical Analysis 2: Comparison: Baloxavir vs Oseltamivir; Day 3; Test type: Superiority; p < 0.0001, van Elteren test — The p-value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 7, analysis 1]
Statistical Analysis 3: Comparison: Baloxavir vs Oseltamivir; Day 4; Test type: Superiority; p = 0.4148, van Elteren test — The p-value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 7, analysis 1]
Statistical Analysis 4: Comparison: Baloxavir vs Oseltamivir; Day 5; Test type: Superiority; p = 0.0338, van Elteren test — The p-value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 7, analysis 1]
Statistical Analysis 5: Comparison: Baloxavir vs Oseltamivir; Day 6; Test type: Superiority; p = 0.9619, van Elteren test — The p-value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 7, analysis 1]
Statistical Analysis 6: Comparison: Baloxavir vs Oseltamivir; Day 9; Test type: Superiority; p = 0.8491, van Elteren test — The p-value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 7, analysis 1]

11. Secondary Outcome: Area Under the Curve (AUC) Adjusted by Baseline in Influenza Virus Titer in Participants Randomized to Baloxavir or Placebo
Description: This endpoint was defined as AUC of change from Baseline in virus titer from Day 1 to Day 9. AUC was calculated using the trapezoidal method.
Time Frame: Day 1 to Day 9
Population: Participants in the intention-to-treat infection population assigned to baloxavir or placebo, with a positive virus titer on Day 1 and available sample on Day 9.
Measure: Mean (Standard Deviation); unit: log₁₀[TCID₅₀/mL]*hours
Arm/Group | Baloxavir | Placebo
Number analyzed (Participants) | 408 | 197
log₁₀[TCID₅₀/mL]*hours | -836.2 (348.9) | -641.8 (377.6)
Statistical Analysis 1: Comparison: Baloxavir vs Placebo; Test type: Superiority; p < 0.0001, van Elteren test — The p-value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 7, analysis 1]

12. Secondary Outcome: Area Under the Curve (AUC) Adjusted by Baseline in Influenza Virus Titer in Adults Randomized to Baloxavir or Oseltamivir
Description: as for outcome 11
Time Frame: Day 1 to Day 9
Population: Participants in the intention-to-treat infection population, ≥ 20 years of age and assigned to baloxavir or oseltamivir, with a positive virus titer on Day 1 and available sample on Day 9.
Measure: Mean (Standard Deviation); unit: log₁₀[TCID₅₀/mL]*hours
Arm/Group | Baloxavir | Oseltamivir
Number analyzed (Participants) | 336 | 340
log₁₀[TCID₅₀/mL]*hours | -829.6 (350.3) | -790.2 (328.4)
Statistical Analysis 1: Comparison: Baloxavir vs Oseltamivir; Test type: Superiority; p = 0.0313, van Elteren test — The p-value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 7, analysis 1]

13. Secondary Outcome: Area Under the Curve (AUC) Adjusted by Baseline of Influenza Virus RNA in Participants Randomized to Baloxavir or Placebo
Description: This endpoint was defined as AUC of change from baseline in the amount of virus RNA (RT-PCR) from Day 1 to Day 9. The AUC was calculated using the trapezoidal method.
Time Frame: Day 1 to Day 9
Population: Participants in the intention-to-treat infection population assigned to baloxavir or placebo with a positive virus RNA determined by RT-PCR at baseline and available sample on Day 9.
Measure: Mean (Standard Deviation); unit: log₁₀ virus particles/mL*hours
Arm/Group | Baloxavir | Placebo
Number analyzed (Participants) | 426 | 208
log₁₀ virus particles/mL*hours | -582.0 (230.9) | -456.8 (269.6)
Statistical Analysis 1: Comparison: Baloxavir vs Placebo; Test type: Superiority; p < 0.0001, van Elteren test — The p-value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 7, analysis 1]

14. Secondary Outcome: Area Under the Curve (AUC) Adjusted by Baseline of Influenza Virus RNA in Adults Randomized to Baloxavir or Oseltamivir
Description: as for outcome 13
Time Frame: Day 1 to Day 9
Population: Participants in the intention-to-treat infection population, ≥ 20 years of age and assigned to baloxavir or oseltamivir, with a positive virus RNA determined by RT-PCR at baseline and available sample on Day 9.
Measure: Mean (Standard Deviation); unit: log₁₀ virus particles/mL*hours
Arm/Group | Baloxavir | Oseltamivir
Number analyzed (Participants) | 351 | 349
log₁₀ virus particles/mL*hours | -581.0 (231.2) | -569.7 (228.8)
Statistical Analysis 1: Comparison: Baloxavir vs Oseltamivir; Test type: Superiority; p = 0.2424, van Elteren test — The p-value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 7, analysis 1]

15. Secondary Outcome: Time to Cessation of Viral Shedding Determined by Virus Titer in Participants Randomized to Baloxavir or Placebo
Description: Time to cessation of viral shedding by virus titer was defined as the time between the initiation of the study treatment and first time when the virus titer was below the limit of detection (0.7 log₁₀[TCID₅₀/mL]). The median and 95% confidence interval (CI) for time to cessation of viral shedding determined by virus titer was analyzed using the Kaplan-Meier (KM) method; participants whose virus titer had not reached cessation by the last observation time point were treated as censored at that time point.
Time Frame: Day 1 to Day 9
Population: Participants in the intention-to-treat infection population assigned to baloxavir or placebo with a positive virus titer on Day 1 whose time to cessation of viral shedding by virus titer was not missing were included in this analysis.
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | Baloxavir | Placebo
Number analyzed (Participants) | 426 | 209
hours | 24.0 [24.0 to 48.0] | 96.0 [NA to NA] — Could not be estimated because lower limit of 95% CI of KM survival function just before the median survival time was higher than 50% and an upper limit of 95% CI of KM survival function just after the median survival time was lower than 50%.
Statistical Analysis 1: Comparison: Baloxavir vs Placebo; Test type: Superiority; p < 0.0001, Generalized Wilcoxon test — The p-value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 1, analysis 1]; Difference = -72.0, 95% CI 2-sided [-72.0 to -48.0]

16. Secondary Outcome: Time to Cessation of Viral Shedding Determined by Virus Titer in Adults Randomized to Baloxavir or Oseltamivir
Description: Time to cessation of viral shedding by virus titer was defined as the time between the initiation of the study treatment and first time when the virus titer was below the limit of detection (0.7 log₁₀[TCID₅₀/mL]). The time to cessation of viral shedding determined by virus titer was analyzed using the Kaplan-Meier (KM) method; participants whose virus titer had not reached cessation by the last observation time point were treated as censored at that time point.
Time Frame: Day 1 to Day 9
Population: Participants in the intention-to-treat infection population, ≥ 20 years of age and assigned to baloxavir or oseltamivir, with a positive virus titer on Day 1 whose time to cessation of viral shedding by virus titer was not missing..
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | Baloxavir | Oseltamivir
Number analyzed (Participants) | 351 | 357
hours | 24.0 [24.0 to 48.0] | 72.0 [72.0 to 96.0]
Statistical Analysis 1: Comparison: Baloxavir vs Oseltamivir; Test type: Superiority; p < 0.0001, Generalized Wilcoxon test — The p-value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 1, analysis 1]; Difference = -48.0, 95% CI 2-sided [-72.0 to -24.0]

17. Secondary Outcome: Time to Cessation of Viral Shedding Determined by Virus RNA in Participants Randomized to Baloxavir or Placebo
Description: Time to cessation of viral shedding by RT-PCR was defined as the time between the initiation of the study treatment and first time when the virus RNA was below the limit of detection measured by RT-PCR.
  Time to cessation of viral shedding by RT-PCR was analyzed using the KM method; participants whose virus RNA had not reached cessation by the last observation time point were treated as censored at that time point.
Time Frame: Day 1 to Day 9
Population: Participants in the intention-to-treat infection population assigned to baloxavir or placebo, with positive influenza virus RNA determined by RT-PCR on Day 1 whose time to cessation of viral shedding by RTPCR was not missing were included in this analysis.
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | Baloxavir | Placebo
Number analyzed (Participants) | 455 | 230
hours | 216.0 [216.0 to 240.0] | 240.0 [240.0 to 336.0]
Statistical Analysis 1: Comparison: Baloxavir vs Placebo; Test type: Superiority; p = 0.0020, Generalized Wilcoxon test — The p-value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 1, analysis 1]; Difference = -24.0, 95% CI 2-sided [-120.0 to 0.0]

18. Secondary Outcome: Time to Cessation of Viral Shedding Determined by Virus RNA in Adults Randomized to Baloxavir or Oseltamivir
Description: as for outcome 17
Time Frame: Day 1 to Day 9
Population: Participants in the intention-to-treat infection population, ≥ 20 years of age and assigned to baloxavir or oseltamivir, with positive influenza virus RNA determined by RT-PCR on Day 1 whose time to cessation of viral shedding by RTPCR was not missing were included in this analysis.
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | Baloxavir | Oseltamivir
Number analyzed (Participants) | 375 | 375
hours | 216.0 [192.0 to 240.0] | 240.0 [216.0 to 240.0]
Statistical Analysis 1: Comparison: Baloxavir vs Oseltamivir; Test type: Superiority; p = 0.0102, Generalized Wilcoxon test — The p-value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 1, analysis 1]; Difference = -24.0, 95% CI 2-sided [-48.0 to 24.0]

19. Secondary Outcome: Percentage of Participants Whose Symptoms Were Alleviated at Each Time Point in Participants Randomized to Baloxavir or Placebo
Description: Participants assessed the severity of seven influenza-associated symptoms (cough, sore throat, headache, nasal congestion, feverishness or chills, muscle or joint pain, and fatigue) on a 4-point scale (with 0 indicating no symptoms, 1 mild symptoms, 2 moderate symptoms, and 3 severe symptoms). Alleviation of symptoms was defined as all seven influenza-related symptoms assessed by the participant as absent (0) or mild (1) .
Time Frame: 12, 24, 36, 48, 72, 96, 120, 144, 168, 192 and 216 hours after the initial dose of study treatment
Population: Participants in the intention-to-treat infection population assigned to baloxavir or placebo with available alleviation of symptoms data at each time point.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Baloxavir | Placebo
Number analyzed (Participants) | 456 | 231
percentage of participants
  12 hours: number analyzed (Participants) | 373 | 197
  12 hours | 9.7 [6.9 to 13.1] | 8.1 [4.7 to 12.9]
  24 hours: number analyzed (Participants) | 445 | 218
  24 hours | 23.1 [19.3 to 27.3] | 12.8 [8.7 to 18.0]
  36 hours: number analyzed (Participants) | 361 | 195
  36 hours | 42.4 [37.2 to 47.7] | 23.1 [17.4 to 29.6]
  48 hours: number analyzed (Participants) | 444 | 220
  48 hours | 50.7 [45.9 to 55.4] | 26.4 [20.7 to 32.7]
  72 hours: number analyzed (Participants) | 431 | 216
  72 hours | 68.9 [64.3 to 73.3] | 49.5 [42.7 to 56.4]
  96 hours: number analyzed (Participants) | 429 | 216
  96 hours | 78.6 [74.4 to 82.3] | 69.9 [63.3 to 75.9]
  120 hours: number analyzed (Participants) | 415 | 212
  120 hours | 85.5 [81.8 to 88.8] | 81.6 [75.7 to 86.6]
  144 hours: number analyzed (Participants) | 404 | 199
  144 hours | 89.1 [85.7 to 92.0] | 85.4 [79.7 to 90.0]
  168 hours: number analyzed (Participants) | 403 | 197
  168 hours | 91.6 [88.4 to 94.1] | 88.3 [83.0 to 92.5]
  192 hours: number analyzed (Participants) | 406 | 197
  192 hours | 90.9 [87.7 to 93.5] | 91.4 [86.5 to 94.9]
  216 hours: number analyzed (Participants) | 224 | 111
  216 hours | 91.1 [86.5 to 94.5] | 91.9 [85.2 to 96.2]
Statistical Analysis 1: Comparison: Baloxavir vs Placebo; 12 hours; Test type: Superiority; p = 0.5973, Mantel Haenszel — The p-value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 3, analysis 1]
Statistical Analysis 2: Comparison: Baloxavir vs Placebo; 24 hours; Test type: Superiority; p = 0.0010, Mantel Haenszel — The p-value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 3, analysis 1]
Statistical Analysis 3: Comparison: Baloxavir vs Placebo; 36 hours; Test type: Superiority; p < 0.0001, Mantel Haenszel — The p-value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 3, analysis 1]
Statistical Analysis 4: Comparison: Baloxavir vs Placebo; 48 hours; Test type: Superiority; p < 0.0001, Mantel Haenszel — The p-value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 3, analysis 1]
Statistical Analysis 5: Comparison: Baloxavir vs Placebo; 72 hours; Test type: Superiority; p < 0.0001, Mantel Haenszel — The p-value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 3, analysis 1]
Statistical Analysis 6: Comparison: Baloxavir vs Placebo; 96 hours; Test type: Superiority; p = 0.0115, Mantel Haenszel — The p-value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 3, analysis 1]
Statistical Analysis 7: Comparison: Baloxavir vs Placebo; 120 hours; Test type: Superiority; p = 0.1298, Mantel Haenszel — The p-value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 3, analysis 1]
Statistical Analysis 8: Comparison: Baloxavir vs Placebo; 144 hours; Test type: Superiority; p = 0.1170, Mantel Haenszel — The p-value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 3, analysis 1]
Statistical Analysis 9: Comparison: Baloxavir vs Placebo; 168 hours; Test type: Superiority; p = 0.0757, Mantel Haenszel — The p-value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 3, analysis 1]
Statistical Analysis 10: Comparison: Baloxavir vs Placebo; 192 hours; Test type: Superiority; p = 0.9453, Mantel Haenszel — The p-value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 3, analysis 1]
Statistical Analysis 11: Comparison: Baloxavir vs Placebo; 216 hours; Test type: Superiority; p = 0.8657, Mantel Haenszel — The p-value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 3, analysis 1]

20. Secondary Outcome: Percentage of Participants Whose Symptoms Were Alleviated at Each Time Point in Adults Randomized to Baloxavir or Oseltamivir
Description: as for outcome 19
Time Frame: 12, 24, 36, 48, 72, 96, 120, 144, 168, 192 and 216 hours after the initial dose of study treatment
Population: Participants in the intention-to-treat infection population, ≥ 20 years of age and assigned to baloxavir or oseltamivir, with available alleviation of symptoms data at each time point.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Baloxavir | Oseltamivir
Number analyzed (Participants) | 376 | 377
percentage of participants
  12 hours: number analyzed (Participants) | 310 | 309
  12 hours | 8.7 [5.8 to 12.4] | 4.9 [2.7 to 7.9]
  24 hours: number analyzed (Participants) | 366 | 365
  24 hours | 21.3 [17.2 to 25.9] | 22.7 [18.5 to 27.4]
  36 hours: number analyzed (Participants) | 299 | 297
  36 hours | 41.1 [35.5 to 46.9] | 38.7 [33.1 to 44.5]
  48 hours: number analyzed (Participants) | 365 | 360
  48 hours | 51.0 [45.7 to 56.2] | 54.4 [49.1 to 59.7]
  72 hours: number analyzed (Participants) | 351 | 359
  72 hours | 70.7 [65.6 to 75.4] | 73.0 [68.1 to 77.5]
  96 hours: number analyzed (Participants) | 351 | 359
  96 hours | 79.8 [75.2 to 83.9] | 80.5 [76.0 to 84.5]
  120 hours: number analyzed (Participants) | 339 | 345
  120 hours | 86.1 [82.0 to 89.6] | 87.0 [82.9 to 90.3]
  144 hours: number analyzed (Participants) | 334 | 334
  144 hours | 89.2 [85.4 to 92.3] | 91.3 [87.8 to 94.1]
  168 hours: number analyzed (Participants) | 336 | 334
  168 hours | 91.4 [87.8 to 94.1] | 94.3 [91.3 to 96.5]
  192 hours: number analyzed (Participants) | 338 | 331
  192 hours | 90.8 [87.2 to 93.7] | 95.5 [92.6 to 97.4]
  216 hours: number analyzed (Participants) | 187 | 188
  216 hours | 90.9 [85.8 to 94.6] | 96.3 [92.5 to 98.5]
Statistical Analysis 1: Comparison: Baloxavir vs Oseltamivir; 12 hours; Test type: Superiority; p = 0.0458, Mantel Haenszel — The p-value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 3, analysis 1]
Statistical Analysis 2: Comparison: Baloxavir vs Oseltamivir; 24 hours; Test type: Superiority; p = 0.7565, Mantel Haenszel — The p-value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 3, analysis 1]
Statistical Analysis 3: Comparison: Baloxavir vs Oseltamivir; 36 hours; Test type: Superiority; p = 0.3297, Mantel Haenszel — The p-value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 3, analysis 1]
Statistical Analysis 4: Comparison: Baloxavir vs Oseltamivir; 48 hours; Test type: Superiority; p = 0.4442, Mantel Haenszel — The p-value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 3, analysis 1]
Statistical Analysis 5: Comparison: Baloxavir vs Oseltamivir; 72 hours; Test type: Superiority; p = 0.6029, Mantel Haenszel — The p-value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 3, analysis 1]
Statistical Analysis 6: Comparison: Baloxavir vs Oseltamivir; 96 hours; Test type: Superiority; p = 0.9881, Mantel Haenszel — The p-value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 3, analysis 1]
Statistical Analysis 7: Comparison: Baloxavir vs Oseltamivir; 120 hours; Test type: Superiority; p = 0.9257, Mantel Haenszel — The p-value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 3, analysis 1]
Statistical Analysis 8: Comparison: Baloxavir vs Oseltamivir; 144 hours; Test type: Superiority; p = 0.5317, Mantel Haenszel — The p-value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 3, analysis 1]
Statistical Analysis 9: Comparison: Baloxavir vs Oseltamivir; 168 hours; Test type: Superiority; p = 0.2144, Mantel Haenszel — The p-value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 3, analysis 1]
Statistical Analysis 10: Comparison: Baloxavir vs Oseltamivir; 192 hours; Test type: Superiority; p = 0.0413, Mantel Haenszel — The p-value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 3, analysis 1]
Statistical Analysis 11: Comparison: Baloxavir vs Oseltamivir; 216 hours; Test type: Superiority; p = 0.0409, Mantel Haenszel — The p-value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 3, analysis 1]

21. Secondary Outcome: Time to Alleviation of the Four Systemic Symptoms in Participants Randomized to Baloxavir or Placebo
Description: Participants assessed the severity of seven influenza-associated symptoms (cough, sore throat, headache, nasal congestion, feverishness or chills, muscle or joint pain, and fatigue) on a 4-point scale (with 0 indicating no symptoms, 1 mild symptoms, 2 moderate symptoms, and 3 severe symptoms).
  Time to alleviation of the 4 systemic symptoms was defined as the time between the initiation of the study treatment to the time when all 4 systemic symptoms (headache, feverishness or chills, muscle or joint pain, and fatigue) were assessed by the participant as 0 (None) or 1 (Mild) for a duration of at least 21.5 hours.
  Time to alleviation of the 4 systemic symptoms was analyzed using KM methods; participants who did not experience alleviation of symptoms were censored at the last observation time point.
Time Frame: Initiation of study treatment up to Day 14
Population: Participants in the intention-to-treat infection population assigned to baloxavir or placebo with available time to alleviation of the 4 systemic symptoms data.
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | Baloxavir | Placebo
Number analyzed (Participants) | 455 | 230
hours | 33.8 [31.0 to 38.3] | 53.5 [45.9 to 57.3]
Statistical Analysis 1: Comparison: Baloxavir vs Placebo; Test type: Superiority; p < 0.0001, Generalized Wilcoxon test — The p-value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 1, analysis 1]; Difference = -19.8

22. Secondary Outcome: Time to Alleviation of the Four Systemic Symptoms in Adults Randomized to Baloxavir or Oseltamivir
Description: as for outcome 21
Time Frame: Initiation of study treatment up to Day 14
Population: Participants in the intention-to-treat infection population, ≥ 20 years of age and assigned to baloxavir or oseltamivir, with available time to alleviation of the 4 systemic symptoms data.
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | Baloxavir | Oseltamivir
Number analyzed (Participants) | 375 | 377
hours | 36.7 [32.0 to 40.1] | 37.4 [31.5 to 42.4]
Statistical Analysis 1: Comparison: Baloxavir vs Oseltamivir; Test type: Superiority; p = 0.4194, Generalized Wilcoxon test — The p-value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 1, analysis 1]; Difference = -0.7

23. Secondary Outcome: Time to Alleviation of the Three Respiratory Symptoms in Participants Randomized to Baloxavir or Placebo
Description: Participants assessed the severity of seven influenza-associated symptoms (cough, sore throat, headache, nasal congestion, feverishness or chills, muscle or joint pain, and fatigue) on a 4-point scale (with 0 indicating no symptoms, 1 mild symptoms, 2 moderate symptoms, and 3 severe symptoms). Time to alleviation of the 3 respiratory symptoms was defined as the time from the start of study treatment to the time when all 3 respiratory symptoms (cough, sore throat and nasal congestion) were assessed by the participant as absent (0) or mild (1) for at least 21.5 hours.
  Time to alleviation of the 3 respiratory symptoms was analyzed using the KM method; participants who did not experience alleviation of symptoms were censored at the last observation time point.
Time Frame: Initiation of study treatment up to Day 14
Population: Participants in the intention-to-treat infection population assigned to baloxavir or placebo with available time to alleviation of the 3 respiratory symptoms data.
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | Baloxavir | Placebo
Number analyzed (Participants) | 455 | 230
hours | 46.0 [43.4 to 50.6] | 69.1 [63.9 to 78.1]
Statistical Analysis 1: Comparison: Baloxavir vs Placebo; Test type: Superiority — The p-value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; p < 0.0001, Generalized Wilcoxon test; [statistical method as in outcome 1, analysis 1]; Difference = -23.1

24. Secondary Outcome: Time to Alleviation of the Three Respiratory Symptoms in Adults Randomized to Baloxavir or Oseltamivir
Description: as for outcome 23
Time Frame: Initiation of study treatment up to Day 14
Population: Participants in the intention-to-treat infection population, ≥ 20 years of age and assigned to baloxavir or oseltamivir, with available time to alleviation of the 3 respiratory symptoms data.
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | Baloxavir | Oseltamivir
Number analyzed (Participants) | 375 | 377
hours | 46.0 [42.7 to 52.0] | 44.6 [40.6 to 49.5]
Statistical Analysis 1: Comparison: Baloxavir vs Oseltamivir; Test type: Superiority; p = 0.4856, Generalized Wilcoxon test — The p-value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 1, analysis 1]; Difference = 1.3

25. Secondary Outcome: Change From Baseline in Composite Symptom Score at Each Time Point in Participants Randomized to Baloxavir or Placebo
Description: Participants assessed the severity of seven influenza-associated symptoms (cough, sore throat, headache, nasal congestion, feverishness or chills, muscle or joint pain, and fatigue) on a 4-point scale (with 0 indicating no symptoms, 1 mild symptoms, 2 moderate symptoms, and 3 severe symptoms).
  The composite symptom score is the total score of the 7 influenza symptoms as assessed by the participant, and ranges from 0 to 21.
Time Frame: Day 1 pretreatment (Baseline) and 12, 24, 36, 48, 72, 96, 120, 144, 168, 192, and 216 hours after the initial dose of study treatment.
Population: Participants in the intention-to-treat infection population assigned to baloxavir or placebo with available composite symptom scores at Baseline and each time point.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Baloxavir | Placebo
Number analyzed (Participants) | 456 | 231
scores on a scale
  12 hours: number analyzed (Participants) | 373 | 197
  12 hours | -2.4 (0.2) | -2.5 (0.3)
  24 hours: number analyzed (Participants) | 445 | 218
  24 hours | -4.7 (0.2) | -3.6 (0.3)
  36 hours: number analyzed (Participants) | 361 | 195
  36 hours | -6.7 (0.2) | -4.9 (0.3)
  48 hours: number analyzed (Participants) | 444 | 220
  48 hours | -7.8 (0.2) | -6.0 (0.3)
  72 hours: number analyzed (Participants) | 431 | 216
  72 hours | -9.4 (0.2) | -8.0 (0.2)
  96 hours: number analyzed (Participants) | 429 | 216
  96 hours | -10.5 (0.2) | -9.5 (0.2)
  120 hours: number analyzed (Participants) | 415 | 212
  120 hours | -10.9 (0.2) | -10.6 (0.2)
  144 hours: number analyzed (Participants) | 404 | 199
  144 hours | -11.6 (0.1) | -11.2 (0.2)
  168 hours: number analyzed (Participants) | 403 | 197
  168 hours | -11.9 (0.1) | -11.8 (0.2)
  192 hours: number analyzed (Participants) | 406 | 197
  192 hours | -12.0 (0.1) | -12.0 (0.2)
  216 hours: number analyzed (Participants) | 224 | 111
  216 hours | -12.4 (0.2) | -12.4 (0.3)
Statistical Analysis 1: Comparison: Baloxavir vs Placebo; 12 hours; Test type: Superiority; p = 0.7173, ANCOVA — The p-value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; Analysis of covariance (ANCOVA) with baseline composite symptom score baseline (≤ 11 or ≥ 12)and region (Japan/Asia, Rest of the world) as covariates; LS Mean Difference = 0.1, 95% CI 2-sided [-0.5 to 0.7], Standard Error of Mean 0.3
Statistical Analysis 2: Comparison: Baloxavir vs Placebo; 24 hours; Test type: Superiority; p = 0.0009, ANCOVA — The p-value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 25, analysis 1]; LS Mean Difference = -1.1, 95% CI 2-sided [-1.7 to -0.4], Standard Error of Mean 0.3
Statistical Analysis 3: Comparison: Baloxavir vs Placebo; 36 hours; Test type: Superiority; p < 0.0001, ANCOVA — The p-value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 25, analysis 1]; LS Mean Difference = -1.8, 95% CI 2-sided [-2.4 to -1.1], Standard Error of Mean 0.3
Statistical Analysis 4: Comparison: Baloxavir vs Placebo; 48 hours; Test type: Superiority; p < 0.0001, ANCOVA — The p-value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 25, analysis 1]; LS Mean Difference = -1.8, 95% CI 2-sided [-2.4 to -1.2], Standard Error of Mean 0.3
Statistical Analysis 5: Comparison: Baloxavir vs Placebo; 72 hours; Test type: Superiority; p < 0.0001, ANCOVA — The p-value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 25, analysis 1]; LS Mean Difference = -1.4, 95% CI 2-sided [-2.0 to -0.9], Standard Error of Mean 0.3
Statistical Analysis 6: Comparison: Baloxavir vs Placebo; 96 hours; Test type: Superiority; p = 0.0001, ANCOVA — The p-value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 25, analysis 1]; LS Mean Difference = -1.0, 95% CI 2-sided [-1.5 to -0.5], Standard Error of Mean 0.3
Statistical Analysis 7: Comparison: Baloxavir vs Placebo; 120 hours; Test type: Superiority; p = 0.1979, ANCOVA — The p-value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 25, analysis 1]; LS Mean Difference = -0.3, 95% CI 2-sided [-0.8 to 0.2], Standard Error of Mean 0.2
Statistical Analysis 8: Comparison: Baloxavir vs Placebo; 144 hours; Test type: Superiority; p = 0.1079, ANCOVA — The p-value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 25, analysis 1]; LS Mean Difference = -0.4, 95% CI 2-sided [-0.8 to 0.1], Standard Error of Mean 0.2
Statistical Analysis 9: Comparison: Baloxavir vs Placebo; 168 hours; Test type: Superiority; p = 0.5805, ANCOVA — The p-value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 25, analysis 1]; LS Mean Difference = -0.1, 95% CI 2-sided [-0.6 to 0.3], Standard Error of Mean 0.2
Statistical Analysis 10: Comparison: Baloxavir vs Placebo; 192 hours; Test type: Superiority; p = 0.8057, ANCOVA — The p-value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 25, analysis 1]; LS Mean Difference = 0.1, 95% CI 2-sided [-0.4 to 0.5], Standard Error of Mean 0.2
Statistical Analysis 11: Comparison: Baloxavir vs Placebo; 216 hours; Test type: Superiority; p = 0.9525, ANCOVA — The p-value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 25, analysis 1]; LS Mean Difference = 0.0, 95% CI 2-sided [-0.6 to 0.6], Standard Error of Mean 0.3

26. Secondary Outcome: Change From Baseline in Composite Symptom Score at Each Time Point in Adults Randomized to Baloxavir or Oseltamivir
Description: as for outcome 25
Time Frame: as for outcome 25
Population: Participants in the intention-to-treat infection population, ≥ 20 years of age and assigned to baloxavir or oseltamivir, with available composite symptom scores at Baseline and each time point.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Baloxavir | Oseltamivir
Number analyzed (Participants) | 376 | 377
scores on a scale
  12 hours: number analyzed (Participants) | 310 | 309
  12 hours | -2.2 (0.2) | -2.4 (0.2)
  24 hours: number analyzed (Participants) | 366 | 365
  24 hours | -4.5 (0.2) | -4.7 (0.2)
  36 hours: number analyzed (Participants) | 299 | 297
  36 hours | -6.5 (0.2) | -6.3 (0.2)
  48 hours: number analyzed (Participants) | 365 | 360
  48 hours | -7.6 (0.2) | -7.8 (0.2)
  72 hours: number analyzed (Participants) | 351 | 359
  72 hours | -9.6 (0.2) | -9.7 (0.2)
  96 hours: number analyzed (Participants) | 351 | 359
  96 hours | -10.5 (0.2) | -10.6 (0.2)
  120 hours: number analyzed (Participants) | 339 | 345
  120 hours | -11.0 (0.2) | -11.3 (0.2)
  144 hours: number analyzed (Participants) | 334 | 334
  144 hours | -11.8 (0.2) | -11.8 (0.2)
  168 hours: number analyzed (Participants) | 336 | 334
  168 hours | -11.9 (0.2) | -12.1 (0.2)
  192 hours: number analyzed (Participants) | 338 | 331
  192 hours | -12.0 (0.1) | -12.4 (0.2)
  216 hours: number analyzed (Participants) | 187 | 188
  216 hours | -12.4 (0.2) | -12.5 (0.2)
Statistical Analysis 1: Comparison: Baloxavir vs Oseltamivir; 12 hours; Test type: Superiority; p = 0.4091, ANCOVA — The p-value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 25, analysis 1]; LS Mean Difference = 0.2, 95% CI 2-sided [-0.3 to 0.8], Standard Error of Mean 0.3
Statistical Analysis 2: Comparison: Baloxavir vs Oseltamivir; 24 hours; Test type: Superiority; p = 0.3073, ANCOVA — The p-value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 25, analysis 1]; LS Mean Difference = 0.3, 95% CI 2-sided [-0.3 to 0.8], Standard Error of Mean 0.3
Statistical Analysis 3: Comparison: Baloxavir vs Oseltamivir; 36 hours; Test type: Superiority; p = 0.3465, ANCOVA — The p-value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 25, analysis 1]; LS Mean Difference = -0.3, 95% CI 2-sided [-0.8 to 0.3], Standard Error of Mean 0.3
Statistical Analysis 4: Comparison: Baloxavir vs Oseltamivir; 48 hours; Test type: Superiority; p = 0.4285, ANCOVA — The p-value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 25, analysis 1]; LS Mean Difference = 0.2, 95% CI 2-sided [-0.3 to 0.7], Standard Error of Mean 0.2
Statistical Analysis 5: Comparison: Baloxavir vs Oseltamivir; 72 hours; Test type: Superiority; p = 0.6703, ANCOVA — The p-value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 25, analysis 1]; LS Mean Difference = 0.1, 95% CI 2-sided [-0.4 to 0.6], Standard Error of Mean 0.2
Statistical Analysis 6: Comparison: Baloxavir vs Oseltamivir; 96 hours; Test type: Superiority; p = 0.7187, ANCOVA — The p-value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 25, analysis 1]; LS Mean Difference = 0.1, 95% CI 2-sided [-0.3 to 0.5], Standard Error of Mean 0.2
Statistical Analysis 7: Comparison: Baloxavir vs Oseltamivir; 120 hours; Test type: Superiority; p = 0.1350, ANCOVA — The p-value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 25, analysis 1]; LS Mean Difference = 0.3, 95% CI 2-sided [-0.1 to 0.7], Standard Error of Mean 0.2
Statistical Analysis 8: Comparison: Baloxavir vs Oseltamivir; 144 hours; Test type: Superiority; p = 0.7046, ANCOVA — The p-value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 25, analysis 1]; LS Mean Difference = 0.1, 95% CI 2-sided [-0.3 to 0.5], Standard Error of Mean 0.2
Statistical Analysis 9: Comparison: Baloxavir vs Oseltamivir; 168 hours; Test type: Superiority; p = 0.2765, ANCOVA — The p-value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 25, analysis 1]; LS Mean Difference = 0.2, 95% CI 2-sided [-0.2 to 0.6], Standard Error of Mean 0.2
Statistical Analysis 10: Comparison: Baloxavir vs Oseltamivir; 192 hours; Test type: Superiority; p = 0.0274, ANCOVA — The p-value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 25, analysis 1]; LS Mean Difference = 0.4, 95% CI 2-sided [0.0 to 0.8], Standard Error of Mean 0.2
Statistical Analysis 11: Comparison: Baloxavir vs Oseltamivir; 216 hours; Test type: Superiority; p = 0.6001, ANCOVA — The p-value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 25, analysis 1]; LS Mean Difference = 0.1, 95% CI 2-sided [-0.3 to 0.6], Standard Error of Mean 0.2

27. Secondary Outcome: Time to Resolution of Fever in Participants Randomized to Baloxavir or Placebo
Description: Time to resolution of fever was defined as the time between the initiation of the study treatment and the resolution of fever. The resolution of fever was defined as the time when the participant's self-measured axillary temperature became less than 37ºC and was maintained at less than 37ºC for a duration of at least 12 hours.
  Time to resolution of fever was analyzed using KM methods; participants who did not experience resolution of fever by the last observation time point were censored at that time point.
Time Frame: Initiation of study treatment up to Day 14
Population: Participants in the intention-to-treat infection population assigned to baloxavir or placebo whose body temperature at baseline was more than 37°C and time to resolution of fever was not missing.
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | Baloxavir | Placebo
Number analyzed (Participants) | 448 | 230
hours | 24.5 [22.6 to 26.6] | 42.0 [37.4 to 44.6]
Statistical Analysis 1: Comparison: Baloxavir vs Placebo; Test type: Superiority; p < 0.0001, Generalized Wilcoxon test — The p-value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 1, analysis 1]; Difference = -17.5, 95% CI 2-sided [-21.1 to -11.9]

28. Secondary Outcome: Time to Resolution of Fever in Adults Randomized to Baloxavir or Oseltamivir
Description: as for outcome 27
Time Frame: Initiation of study treatment up to Day 14
Population: Participants in the intention-to-treat infection population, ≥ 20 years of age and assigned to baloxavir or oseltamivir, whose body temperature at baseline was more than 37°C and time to resolution of fever was not missing.
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | Baloxavir | Oseltamivir
Number analyzed (Participants) | 369 | 374
hours | 24.4 [22.2 to 26.5] | 24.0 [22.1 to 25.9]
Statistical Analysis 1: Comparison: Baloxavir vs Oseltamivir; Test type: Superiority; p = 0.9225, Generalized Wilcoxon test — The p-value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 1, analysis 1]

29. Secondary Outcome: Percentage of Participants Reporting Normal Temperature at Each Time Point in Participants Randomized to Baloxavir or Placebo
Description: Defined as the percentage of patients whose axillary temperature dropped to less than 37ºC after the initiation of study treatment.
Time Frame: 12, 24, 36, 48, 72, 96, 120, 144, 168, 192 and 216 hours after the initial dose of study treatment
Population: Participants in the intention-to-treat infection population assigned to baloxavir or placebo whose body temperature at baseline was more than 37°C with available body temperature data at each time point.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Baloxavir | Placebo
Number analyzed (Participants) | 449 | 230
percentage of participants
  12 hours: number analyzed (Participants) | 431 | 217
  12 hours | 26.5 [22.3 to 30.9] | 25.3 [19.7 to 31.7]
  24 hours: number analyzed (Participants) | 442 | 225
  24 hours | 64.3 [59.6 to 68.7] | 48.4 [41.8 to 55.2]
  36 hours: number analyzed (Participants) | 428 | 218
  36 hours | 80.8 [76.8 to 84.5] | 58.3 [51.4 to 64.9]
  48 hours: number analyzed (Participants) | 439 | 220
  48 hours | 89.3 [86.0 to 92.0] | 67.3 [60.6 to 73.4]
  72 hours: number analyzed (Participants) | 413 | 197
  72 hours | 93.7 [90.9 to 95.8] | 83.8 [77.8 to 88.6]
  96 hours: number analyzed (Participants) | 400 | 197
  96 hours | 92.8 [89.8 to 95.1] | 93.9 [89.6 to 96.8]
  120 hours: number analyzed (Participants) | 392 | 194
  120 hours | 92.9 [89.8 to 95.2] | 92.8 [88.2 to 96.0]
  144 hours: number analyzed (Participants) | 379 | 187
  144 hours | 93.4 [90.4 to 95.7] | 93.6 [89.1 to 96.6]
  168 hours: number analyzed (Participants) | 375 | 187
  168 hours | 93.3 [90.3 to 95.6] | 93.6 [89.1 to 96.6]
  192 hours: number analyzed (Participants) | 374 | 191
  192 hours | 94.1 [91.2 to 96.3] | 93.7 [89.3 to 96.7]
  216 hours: number analyzed (Participants) | 372 | 191
  216 hours | 92.5 [89.3 to 94.9] | 92.7 [88.0 to 95.9]
Statistical Analysis 1: Comparison: Baloxavir vs Placebo; 12 hours; Test type: Superiority; p = 0.7866, Mantel Haenszel — The p-value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 3, analysis 1]
Statistical Analysis 2: Comparison: Baloxavir vs Placebo; 24 hours; Test type: Superiority; p < 0.0001, Mantel Haenszel — The p-value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 3, analysis 1]
Statistical Analysis 3: Comparison: Baloxavir vs Placebo; 36 hours; Test type: Superiority; p < 0.0001, Mantel Haenszel — The p-value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 3, analysis 1]
Statistical Analysis 4: Comparison: Baloxavir vs Placebo; 48 hours; Test type: Superiority; p < 0.0001, Mantel Haenszel — The p-value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 3, analysis 1]
Statistical Analysis 5: Comparison: Baloxavir vs Placebo; 72 hours; Test type: Superiority; p < 0.0001, Mantel Haenszel — The p-value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 3, analysis 1]
Statistical Analysis 6: Comparison: Baloxavir vs Placebo; 96 hours; Test type: Superiority; p = 0.7044, Mantel Haenszel — The p-value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 3, analysis 1]
Statistical Analysis 7: Comparison: Baloxavir vs Placebo; 120 hours; Test type: Superiority; p = 0.8512, Mantel Haenszel — The p-value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 3, analysis 1]
Statistical Analysis 8: Comparison: Baloxavir vs Placebo; 144 hours; Test type: Superiority; p = 0.8783, Mantel Haenszel — The p-value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 3, analysis 1]
Statistical Analysis 9: Comparison: Baloxavir vs Placebo; 168 hours; Test type: Superiority; p = 0.8291, Mantel Haenszel — The p-value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 3, analysis 1]
Statistical Analysis 10: Comparison: Baloxavir vs Placebo; 192 hours; Test type: Superiority; p = 0.8644, Mantel Haenszel — The p-value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 3, analysis 1]
Statistical Analysis 11: Comparison: Baloxavir vs Placebo; 216 hours; Test type: Superiority; p = 0.9312, Mantel Haenszel — The p-value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 3, analysis 1]

30. Secondary Outcome: Percentage of Participants Reporting Normal Temperature at Each Time Point in Adults Randomized to Baloxavir or Oseltamivir
Description: as for outcome 29
Time Frame: 12, 24, 36, 48, 72, 96, 120, 144, 168, 192 and 216 hours after the initial dose of study treatment
Population: Participants in the intention-to-treat infection population, ≥ 20 years of age and assigned to baloxavir or oseltamivir, whose body temperature at baseline was more than 37°C with available body temperature data at each time point.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Baloxavir | Oseltamivir
Number analyzed (Participants) | 370 | 374
percentage of participants
  12 hours: number analyzed (Participants) | 360 | 353
  12 hours | 25.0 [20.6 to 29.8] | 28.3 [23.7 to 33.3]
  24 hours: number analyzed (Participants) | 364 | 367
  24 hours | 64.3 [59.1 to 69.2] | 66.8 [61.7 to 71.6]
  36 hours: number analyzed (Participants) | 354 | 359
  36 hours | 81.9 [77.5 to 85.8] | 79.1 [74.5 to 83.2]
  48 hours: number analyzed (Participants) | 363 | 366
  48 hours | 90.1 [86.5 to 93.0] | 89.9 [86.3 to 92.8]
  72 hours: number analyzed (Participants) | 339 | 344
  72 hours | 93.8 [90.7 to 96.1] | 89.5 [85.8 to 92.6]
  96 hours: number analyzed (Participants) | 329 | 334
  96 hours | 93.9 [90.8 to 96.2] | 94.9 [92.0 to 97.0]
  120 hours: number analyzed (Participants) | 324 | 335
  120 hours | 93.8 [90.6 to 96.2] | 95.8 [93.1 to 97.7]
  144 hours: number analyzed (Participants) | 320 | 328
  144 hours | 92.8 [89.4 to 95.4] | 94.5 [91.5 to 96.7]
  168 hours: number analyzed (Participants) | 314 | 315
  168 hours | 93.6 [90.3 to 96.1] | 95.9 [93.0 to 97.8]
  192 hours: number analyzed (Participants) | 313 | 308
  192 hours | 94.6 [91.4 to 96.8] | 95.8 [92.9 to 97.7]
  216 hours: number analyzed (Participants) | 305 | 309
  216 hours | 92.8 [89.3 to 95.4] | 94.5 [91.3 to 96.8]
Statistical Analysis 1: Comparison: Baloxavir vs Oseltamivir; 12 hours; Test type: Superiority; p = 0.2953, Mantel Haenszel — The p-value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 3, analysis 1]
Statistical Analysis 2: Comparison: Baloxavir vs Oseltamivir; 24 hours; Test type: Superiority; p = 0.5414, Mantel Haenszel — The p-value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 3, analysis 1]
Statistical Analysis 3: Comparison: Baloxavir vs Oseltamivir; 36 hours; Test type: Superiority; p = 0.2079, Mantel Haenszel — The p-value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 3, analysis 1]
Statistical Analysis 4: Comparison: Baloxavir vs Oseltamivir; 48 hours; Test type: Superiority; p = 0.7771, Mantel Haenszel — The p-value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 3, analysis 1]
Statistical Analysis 5: Comparison: Baloxavir vs Oseltamivir; 72 hours; Test type: Superiority; p = 0.0215, Mantel Haenszel — The p-value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 3, analysis 1]
Statistical Analysis 6: Comparison: Baloxavir vs Oseltamivir; 96 hours; Test type: Superiority; p = 0.8033, Mantel Haenszel — The p-value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 3, analysis 1]
Statistical Analysis 7: Comparison: Baloxavir vs Oseltamivir; 120 hours; Test type: Superiority; p = 0.4157, Mantel Haenszel — The p-value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 3, analysis 1]
Statistical Analysis 8: Comparison: Baloxavir vs Oseltamivir; 144 hours; Test type: Superiority; p = 0.5908, Mantel Haenszel — The p-value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 3, analysis 1]
Statistical Analysis 9: Comparison: Baloxavir vs Oseltamivir; 168 hours; Test type: Superiority; p = 0.2975, Mantel Haenszel — The p-value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 3, analysis 1]
Statistical Analysis 10: Comparison: Baloxavir vs Oseltamivir; 192 hours; Test type: Superiority; p = 0.8644, Mantel Haenszel — The p-value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 3, analysis 1]
Statistical Analysis 11: Comparison: Baloxavir vs Oseltamivir; 216 hours; Test type: Superiority; p = 0.5573, Mantel Haenszel — The p-value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05.m; [statistical method as in outcome 3, analysis 1]

31. Secondary Outcome: Body Temperature at Each Time Point in Participants Randomized to Baloxavir or Placebo
Description: Participant's self-measured axillary temperature using an electronic thermometer.
Time Frame: 12, 24, 36, 48, 72, 96 and 120 hours after the initial dose of study treatment
Population: Participants in the intention-to-treat infection population assigned to baloxavir or placebo with available temperature data at each time point.
Measure: Least Squares Mean (Standard Error); unit: °C
Arm/Group | Baloxavir | Placebo
Number analyzed (Participants) | 456 | 231
°C
  12 hours: number analyzed (Participants) | 435 | 218
  12 hours | 37.40 (0.05) | 37.49 (0.07)
  24 hours: number analyzed (Participants) | 447 | 226
  24 hours | 36.73 (0.04) | 37.07 (0.05)
  36 hours: number analyzed (Participants) | 432 | 219
  36 hours | 36.49 (0.04) | 36.90 (0.05)
  48 hours: number analyzed (Participants) | 446 | 221
  48 hours | 36.32 (0.03) | 36.69 (0.05)
  72 hours: number analyzed (Participants) | 418 | 198
  72 hours | 36.26 (0.03) | 36.48 (0.04)
  96 hours: number analyzed (Participants) | 405 | 198
  96 hours | 36.27 (0.03) | 36.31 (0.04)
  120 hours: number analyzed (Participants) | 396 | 195
  120 hours | 36.28 (0.03) | 36.25 (0.04)
Statistical Analysis 1: Comparison: Baloxavir vs Placebo; 12 hours; Test type: Superiority; p = 0.2557, ANCOVA — The p-value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; ANCOVA with baseline composite symptom score and region (Japan/Asia, Rest of the world) and body temperature at baseline as covariates; LS Mean Difference = -0.09, 95% CI 2-sided [-0.24 to 0.06], Standard Error of Mean 0.08
Statistical Analysis 2: Comparison: Baloxavir vs Placebo; 24 hours; Test type: Superiority; p < 0.0001, ANCOVA — The p-value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 31, analysis 1]; LS Mean Difference = -0.34, 95% CI 2-sided [-0.46 to -0.22], Standard Error of Mean 0.06
Statistical Analysis 3: Comparison: Baloxavir vs Placebo; 36 hours; Test type: Superiority; p < 0.0001, ANCOVA — The p-value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 31, analysis 1]; LS Mean Difference = -0.41, 95% CI 2-sided [-0.52 to -0.29], Standard Error of Mean 0.06
Statistical Analysis 4: Comparison: Baloxavir vs Placebo; 48 hours; Test type: Superiority; p < 0.0001, ANCOVA — The p-value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 31, analysis 1]; LS Mean Difference = -0.37, 95% CI 2-sided [-0.48 to -0.27], Standard Error of Mean 0.05
Statistical Analysis 5: Comparison: Baloxavir vs Placebo; 72 hours; Test type: Superiority; p < 0.0001, ANCOVA — The p-value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 31, analysis 1]; LS Mean Difference = -0.22, 95% CI 2-sided [-0.31 to -0.13], Standard Error of Mean 0.05
Statistical Analysis 6: Comparison: Baloxavir vs Placebo; 96 hours; Test type: Superiority; p = 0.4484, ANCOVA — The p-value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 31, analysis 1]; LS Mean Dfference = -0.04, 95% CI 2-sided [-0.13 to 0.06], Standard Error of Mean 0.05
Statistical Analysis 7: Comparison: Baloxavir vs Placebo; ANCOVA with baseline composite symptom score and region (Japan/Asia, Rest of the world) and body temperature at baseline as covariates; Test type: Superiority; p = 0.5963, ANCOVA — The p-value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 31, analysis 1]; LS Mean Difference = 0.02, 95% CI 2-sided [-0.07 to 0.11], Standard Error of Mean 0.05

32. Secondary Outcome: Body Temperature at Each Time Point in Adults Randomized to Baloxavir or Oseltamivir
Description: Participant's self-measured axillary temperature using an electronic thermometer.
Time Frame: 12, 24, 36, 48, 72, 96 and 120 hours after the initial dose of study treatment
Population: Participants in the intention-to-treat infection population, ≥ 20 years of age and assigned to baloxavir or oseltamivir, with available temperature data at each time point.
Measure: Least Squares Mean (Standard Error); unit: °C
Arm/Group | Baloxavir | Oseltamivir
Number analyzed (Participants) | 376 | 377
°C
  12 hours: number analyzed (Participants) | 363 | 355
  12 hours | 37.47 (0.05) | 37.35 (0.05)
  24 hours: number analyzed (Participants) | 368 | 369
  24 hours | 36.78 (0.04) | 36.73 (0.04)
  36 hours: number analyzed (Participants) | 358 | 362
  36 hours | 36.55 (0.04) | 36.54 (0.04)
  48 hours: number analyzed (Participants) | 369 | 369
  48 hours | 36.34 (0.03) | 36.36 (0.03)
  72 hours: number analyzed (Participants) | 344 | 346
  72 hours | 36.30 (0.03) | 36.31 (0.03)
  96 hours: number analyzed (Participants) | 334 | 337
  96 hours | 36.26 (0.03) | 36.23 (0.03)
  120 hours: number analyzed (Participants) | 328 | 337
  120 hours | 36.27 (0.03) | 36.21 (0.03)
Statistical Analysis 1: Comparison: Baloxavir vs Oseltamivir; 12 hours; Test type: Superiority; p = 0.0937, ANCOVA — The p-value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 31, analysis 1]; LS Mean Difference = 0.11, 95% CI 2-sided [-0.02 to 0.24], Standard Error of Mean 0.07
Statistical Analysis 2: Comparison: Baloxavir vs Oseltamivir; 24 hours; Test type: Superiority; p = 0.3343, ANCOVA — The p-value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 31, analysis 1]; LS Mean Difference = 0.05, 95% CI 2-sided [-0.05 to 0.16], Standard Error of Mean 0.05
Statistical Analysis 3: Comparison: Baloxavir vs Oseltamivir; 36 hours; Test type: Superiority; p = 0.9258, ANCOVA — The p-value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 31, analysis 1]; LS Mean Difference = 0.00, 95% CI 2-sided [-0.09 to 0.10], Standard Error of Mean 0.05
Statistical Analysis 4: Comparison: Baloxavir vs Oseltamivir; 48 hours; Test type: Superiority; p = 0.6574, ANCOVA — The p-value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 31, analysis 1]; LS Mean Difference = -0.02, 95% CI 2-sided [-0.10 to 0.06], Standard Error of Mean 0.04
Statistical Analysis 5: Comparison: Baloxavir vs Oseltamivir; 72 hours; Test type: Superiority; p = 0.8520, ANCOVA — The p-value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 31, analysis 1]; LS Mean Difference = -0.01, 95% CI 2-sided [-0.09 to 0.07], Standard Error of Mean 0.04
Statistical Analysis 6: Comparison: Baloxavir vs Oseltamivir; 96 hours; Test type: Superiority; p = 0.4532, ANCOVA — The p-value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 31, analysis 1]; LS Mean Difference = 0.03, 95% CI 2-sided [-0.05 to 0.11], Standard Error of Mean 0.04
Statistical Analysis 7: Comparison: Baloxavir vs Oseltamivir; 120 hours; Test type: Superiority; p = 0.1570, ANCOVA — The p-value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 31, analysis 1]; LS Mean Difference = 0.05, 95% CI 2-sided [-0.02 to 0.13], Standard Error of Mean 0.04

33. Secondary Outcome: Time to Alleviation of Individual Symptoms in Participants Randomized to Baloxavir or Placebo
Description: Participants assessed the severity of seven influenza-associated symptoms (cough, sore throat, headache, nasal congestion, feverishness or chills, muscle or joint pain, and fatigue) on a 4-point scale (with 0 indicating no symptoms, 1 mild symptoms, 2 moderate symptoms, and 3 severe symptoms).
  Time to alleviation of each symptom was defined as the time from the start of treatment to the start of the time period when the individual symptom was assessed by the participant as 0 (None) or 1 (Mild) for a duration of at least 21.5 hours.
Time Frame: Initiation of study treatment up to Day 14
Population: Participants in the intention-to-treat infection population assigned to baloxavir or placebo whose symptom score at baseline was moderate (2) or severe (3) with available time to alleviation of symptoms data.
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | Baloxavir | Placebo
Number analyzed (Participants) | 455 | 230
hours
  Cough: number analyzed (Participants) | 308 | 171
  Cough | 38.3 [30.3 to 43.5] | 61.4 [44.8 to 69.5]
  Sore Throat: number analyzed (Participants) | 249 | 119
  Sore Throat | 31.5 [27.3 to 39.2] | 40.5 [31.8 to 48.3]
  Headache: number analyzed (Participants) | 296 | 153
  Headache | 26.1 [22.9 to 29.8] | 37.9 [25.8 to 42.2]
  Nasal Congestion: number analyzed (Participants) | 277 | 153
  Nasal Congestion | 31.8 [29.9 to 38.7] | 52.5 [41.5 to 62.7]
  Feverishness or chills: number analyzed (Participants) | 408 | 214
  Feverishness or chills | 20.9 [20.0 to 21.9] | 25.8 [21.7 to 31.5]
  Muscle or joint pain: number analyzed (Participants) | 353 | 169
  Muscle or joint pain | 23.2 [21.4 to 26.3] | 31.3 [25.5 to 39.2]
  Fatigue: number analyzed (Participants) | 361 | 188
  Fatigue | 25.3 [22.0 to 29.2] | 40.5 [31.2 to 46.8]
Statistical Analysis 1: Comparison: Baloxavir vs Placebo; Cough; Test type: Superiority; p = 0.0001, Generalized Wilcoxon test — The p-value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 1, analysis 1]; Difference = -23.1
Statistical Analysis 2: Comparison: Baloxavir vs Placebo; Sore throat; Test type: Superiority; p = 0.0298, Generalized Wilcoxon test — The p-value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 1, analysis 1]; Difference = -9.0
Statistical Analysis 3: Comparison: Baloxavir vs Placebo; Headache; Test type: Superiority; p = 0.0297, Generalized Wilcoxon test — The p-value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 1, analysis 1]; Difference = -11.8
Statistical Analysis 4: Comparison: Baloxavir vs Placebo; Nasal Congestion; Test type: Superiority; p = 0.0027, Generalized Wilcoxon test — The p-value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 1, analysis 1]; Difference = -20.7
Statistical Analysis 5: Comparison: Baloxavir vs Placebo; Feverishness or chills; Test type: Superiority; p = 0.0003, Generalized Wilcoxon test — The p-value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 1, analysis 1]; Difference = -4.9
Statistical Analysis 6: Comparison: Baloxavir vs Placebo; Muscle or joint pain; Test type: Superiority; p = 0.0094, Generalized Wilcoxon test — The p-value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 1, analysis 1]; Difference = -8.1
Statistical Analysis 7: Comparison: Baloxavir vs Placebo; Fatigue; Test type: Superiority; p = 0.0007, Generalized Wilcoxon test — The p-value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 1, analysis 1]; Difference = -15.3

34. Secondary Outcome: Time to Alleviation of Individual Symptoms in Adults Randomized to Baloxavir or Oseltamivir
Description: as for outcome 33
Time Frame: Initiation of study treatment up to Day 14
Population: Participants in the intention-to-treat infection population, ≥ 20 years of age and assigned to baloxavir or oseltamivir, whose symptom score at baseline was moderate (2) or severe (3) with available time to alleviation of symptoms data.
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | Baloxavir | Oseltamivir
Number analyzed (Participants) | 375 | 377
hours
  Cough: number analyzed (Participants) | 250 | 262
  Cough | 38.2 [30.3 to 43.4] | 31.4 [28.6 to 36.8]
  Sore Throat: number analyzed (Participants) | 211 | 198
  Sore Throat | 32.1 [27.6 to 39.8] | 30.4 [25.0 to 43.9]
  Headache: number analyzed (Participants) | 246 | 239
  Headache | 26.9 [24.5 to 30.8] | 25.6 [21.9 to 30.4]
  Nasal Congestion: number analyzed (Participants) | 217 | 230
  Nasal Congestion | 33.0 [30.5 to 40.4] | 31.3 [26.8 to 39.8]
  Feverishness or chills: number analyzed (Participants) | 337 | 341
  Feverishness or chills | 21.0 [20.0 to 22.0] | 21.2 [20.3 to 22.0]
  Muscle or joint pain: number analyzed (Participants) | 300 | 291
  Muscle or joint pain | 23.3 [21.6 to 26.7] | 24.0 [21.6 to 27.1]
  Fatigue: number analyzed (Participants) | 293 | 308
  Fatigue | 28.9 [23.2 to 30.5] | 26.6 [23.0 to 30.8]
Statistical Analysis 1: Comparison: Baloxavir vs Oseltamivir; Cough; Test type: Superiority; p = 0.6623, Generalized Wilcoxon test — The p-value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 1, analysis 1]; Difference = 6.8
Statistical Analysis 2: Comparison: Baloxavir vs Oseltamivir; Sore throat; Test type: Superiority; p = 0.8184, Generalized Wilcoxon test — The p-value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 1, analysis 1]; Difference = 1.8
Statistical Analysis 3: Comparison: Baloxavir vs Oseltamivir; Headache; Test type: Superiority; p = 0.9989, Generalized Wilcoxon test — The p-value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 1, analysis 1]; Difference = 1.3
Statistical Analysis 4: Comparison: Baloxavir vs Oseltamivir; Nasal congestion; Test type: Superiority; p = 0.3706, Generalized Wilcoxon test — The p-value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 1, analysis 1]; Difference = 1.7
Statistical Analysis 5: Comparison: Baloxavir vs Oseltamivir; Feverishness or chills; Test type: Superiority; p = 0.9973, Generalized Wilcoxon test — The p-value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 1, analysis 1]; Difference = -0.1
Statistical Analysis 6: Comparison: Baloxavir vs Oseltamivir; Muscle or joint pain; Test type: Superiority; p = 0.6760, Generalized Wilcoxon test — The p-value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 1, analysis 1]; Difference = -0.7
Statistical Analysis 7: Comparison: Baloxavir vs Oseltamivir; Fatigue; Test type: Superiority; p = 0.4241, Generalized Wilcoxon test — The p-value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 1, analysis 1]; Difference = 2.2

35. Secondary Outcome: Time to Return to Preinfluenza Health Status in Participants Randomized to Baloxavir or Placebo
Description: Participants were asked to record their preinfluenza health status on a scale from 0 (worst possible health) to 10 (normal health [for someone your age and your health condition]), and their health status every day after initiation of study treatment on the same scale. Return to preinfluenza health status was defined as time from the initiation of the study treatment to the first time when the health status score was equal to or higher than the preinfluenza health status score.
  Time to return to preinfluenza health status was analyzed using KM methods; participants with a smaller number on the scale for health status by the last observation time point were censored at that time point.
Time Frame: Initiation of study treatment up to Day 14
Population: Participants in the intention-to-treat infection population assigned to baloxavir or placebo whose health status score at baseline was lower than the preinfluenza health status score and with available time to return to preinfluenza health status data.
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | Baloxavir | Placebo
Number analyzed (Participants) | 378 | 190
hours | 129.2 [122.1 to 152.3] | 168.8 [145.9 to 202.2]
Statistical Analysis 1: Comparison: Baloxavir vs Placebo; Test type: Superiority — The p-value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; p = 0.0563, Generalized Wilcoxon test; [statistical method as in outcome 1, analysis 1]; Difference = -39.5

36. Secondary Outcome: Time to Return to Preinfluenza Health Status in Adults Randomized to Baloxavir or Oseltamivir
Description: as for outcome 35
Time Frame: Initiation of study treatment up to Day 14
Population: Participants in the intention-to-treat infection population, ≥ 20 years of age and assigned to baloxavir or oseltamivir, whose health status score at baseline was lower than the preinfluenza health status score and with available time to return to preinfluenza health status data.
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | Baloxavir | Oseltamivir
Number analyzed (Participants) | 314 | 308
hours | 127.8 [121.5 to 152.8] | 128.5 [122.8 to 151.0]
Statistical Analysis 1: Comparison: Baloxavir vs Oseltamivir; Test type: Superiority; p = 0.7176, Generalized Wilcoxon test — The p-value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 1, analysis 1]; Difference = -0.6

37. Secondary Outcome: Percentage of Participants With Influenza-related Complications in Participants Randomized to Baloxavir or Placebo
Description: The percentage of participants who experienced each influenza-related complication (hospitalization, death, sinusitis, otitis media, bronchitis, and radiologically confirmed pneumonia) as an adverse event after the initiation of the study treatment.
Time Frame: Initiation of study treatment up to Day 14
Population: Participants in the intention-to-treat infection population assigned to baloxavir or placebo
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Baloxavir | Placebo
Number analyzed (Participants) | 456 | 231
percentage of participants
  Any complication | 3.5 [2.0 to 5.6] | 4.3 [2.1 to 7.8]
  Death | 0 [0.0 to 0.8] | 0 [0.0 to 1.6]
  Hospitalization | 0 [0.0 to 0.8] | 0 [0.0 to 1.6]
  Sinusitis | 0.9 [0.2 to 2.2] | 0.9 [0.1 to 3.1]
  Otitis media | 0.4 [0.1 to 1.6] | 0 [0.0 to 1.6]
  Bronchitis | 2.0 [0.9 to 3.7] | 3.5 [1.5 to 6.7]
  Pneumonia | 0.4 [0.1 to 1.6] | 0.4 [0.0 to 2.4]
Statistical Analysis 1: Comparison: Baloxavir vs Placebo; Any Complications; Test type: Superiority; p = 0.6728, Fisher Exact — The p-value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05

38. Secondary Outcome: Percentage of Participants With Influenza-related Complications in Adults Randomized to Baloxavir or Oseltamivir
Description: as for outcome 37
Time Frame: Initiation of study treatment up to Day 14
Population: Participants in the intention-to-treat infection population ≥ 20 years of age and assigned to baloxavir or oseltamivir.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Baloxavir | Oseltamivir
Number analyzed (Participants) | 376 | 377
percentage of participants
  Any complication | 4.0 [2.2 to 6.5] | 2.4 [1.1 to 4.5]
  Death | 0 [0.0 to 1.0] | 0 [0.0 to 1.0]
  Hospitalization | 0 [0.0 to 1.0] | 0.3 [0.0 to 1.5]
  Sinusitis | 0.8 [0.2 to 2.3] | 0 [0.0 to 1.0]
  Otitis media | 0.5 [0.1 to 1.9] | 0.3 [0.0 to 1.5]
  Bronchitis | 2.4 [1.1 to 4.5] | 1.6 [0.6 to 3.4]
  Pneumonia | 0.5 [0.1 to 1.9] | 0.3 [0.0 to 1.5]
Statistical Analysis 1: Comparison: Baloxavir vs Oseltamivir; Any Complications; Test type: Superiority; p = 0.2217, Fisher Exact — The p-value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05

39. Secondary Outcome: Percentage of Participants With Adverse Events (AEs)
Time Frame: From first dose of study drug to Day 22
Population: All participants who received at least 1 dose of study drug
Measure: Number; unit: percentage of participants
Arm/Group | Baloxavir | Placebo | Oseltamivir
Number analyzed (Participants) | 610 | 309 | 513
percentage of participants
  Adverse events (AEs) | 20.7 | 24.6 | 24.8
  Serious adverse events (SAEs) | 0.3 | 0.0 | 0.0
  AEs leading to withdrawal of study drug | 0.3 | 0.3 | 0.4
  Treatment-related adverse events (TRAEs) | 4.4 | 3.9 | 8.4
  Treatment-related serious adverse events | 0.0 | 0.0 | 0.0
  TRAEs leading to withdrawal of study drug | 0.0 | 0.3 | 0.2

ADVERSE EVENTS:
Time Frame: From first dose of treatment to Day 22
Arm/Group | Baloxavir | Placebo | Oseltamivir
All-Cause Mortality (participants affected / at risk) | 0/610 | 0/309 | 0/513
Serious Adverse Events (participants affected / at risk) | 2/610 | 0/309 | 0/513
Other Adverse Events (participants affected / at risk) | 47/610 | 40/309 | 45/513
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Baloxavir (N=610) | Placebo (N=309) | Oseltamivir (N=513)
Meningitis viral (Infections and infestations) | 1 | 0 | 0
Incarcerated inguinal hernia (Gastrointestinal disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Baloxavir (N=610) | Placebo (N=309) | Oseltamivir (N=513)
Bronchitis (Infections and infestations) | 16 | 17 | 18
Sinusitis (Infections and infestations) | 7 | 8 | 5
Diarrhoea (Gastrointestinal disorders) | 18 | 14 | 11
Nausea (Gastrointestinal disorders) | 8 | 4 | 16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can embargo results from a PI's center until the combined results from the completed study have been published in full or the sponsor confirms there will be no multicenter study publication. Results communications must be provided to the sponsor for review at least 60 days before submission for publication. By written request, the sponsor can extend the embargo up to an additional 60 days. The sponsor cannot require changes to scientific content and cannot further extend the embargo.

DOCUMENTS (2):
  • Study Protocol (2016-10-31): https://cdn.clinicaltrials.gov/large-docs/54/NCT02954354/Prot_000.pdf
  • Statistical Analysis Plan (2017-07-06): https://cdn.clinicaltrials.gov/large-docs/54/NCT02954354/SAP_001.pdf